CLINICAL TRIAL: NCT03613649
Title: A Phase 1, Randomized, Double-blinded, Four-period Crossover, Thorough QT/QTC (TQT) Clinical Trial to Evaluate the Effect of Zoliflodacin on Cardiac Repolarization in Healthy Male and Female Subjects
Brief Title: Thorough QT/QTC (TQT) Clinical Trial to Evaluate the Effect of Zoliflodacin on Cardiac Repolarization in Healthy Male and Female Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 16-0110; HHSN272201500005I
Record Dates: First submitted 2018-07-26; First posted 2018-08-03 (Actual); Results first posted 2020-03-27 (Actual); Last update posted 2020-03-27 (Actual); Status verified 2019-05-07

CONDITIONS: Electrocardiogram Repolarisation Abnormality; Gonococcal Infection
Keywords: AZD0914; Cardiac; ETX0914; Healthy; Moxifloxacin; Repolarization; Study; TQT; Volunteers; Zoliflodacin
MeSH Terms: conditions — Gonorrhea | interventions — zoliflodacin; Moxifloxacin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Treatment A (Experimental): 2 g of zoliflodacin administered orally on Day 1 of each dosing period, n=72
  Interventions: Drug: AZD0914
- Treatment B (Experimental): 4 g of zoliflodacin administered orally on Day 1 of each dosing period, n=72
  Interventions: Drug: AZD0914
- Treatment C (Placebo Comparator): Placebo for zoliflodacin administered orally on Day 1 of each dosing period, n=72
  Interventions: Other: Placebo
- Treatment D (Active Comparator): 400 mg of moxifloxacin administered orally on Day 1 of each dosing period, n=72
  Interventions: Drug: Moxifloxacin

INTERVENTIONS:
Drug: AZD0914 — Spiropyrimidinetrione antibacterial drug, which inhibits bacterial DNA synthesis by a novel mechanism. Powder will be reconstituted in 60 mL of tap water and dosed orally after an overnight fast. After the cup containing 60 mL of zoliflodacin is taken, approximately 60 mL of tap water will be added to the cup and consumed by the subject to chase the initial dose.
  Arms: Treatment A; Treatment B
Drug: Moxifloxacin — Broad-spectrum 8-methoxy fluoroquinolone with activity against both Gram-positive and Gram-negative bacteria, including anaerobes. A single, commercially-available, film-coated, 400-mg tablet of moxifloxacin hydrochloride will be administered orally with 120 mL of tap water.
  Arms: Treatment D
Other: Placebo — Composed of 4 g of the same excipients found in zoliflodacin. Powder will be reconstituted in 60 mL of tap water and dosed orally after an overnight fast. After the cup containing 60 mL of placebo is taken, approximately 60 mL of tap water will be added to the cup and consumed by the subject to chase the initial dose.
  Arms: Treatment C

SUMMARY:
The Phase I Thorough QT/QTc (TQT) study will be performed in a single center, the Vince & Associates Clinical Research, Inc., clinical trials unit (CTU), in 72 healthy male or female subjects, aged 18 to 45 years inclusive, to evaluate the effect of zoliflodacin on the corrected QT interval of the electrocardiogram (ECG) using Fridericia's Formula (QTcF) and other ECG parameters; the correlation of the drug concentrations (and pharmacokinetic (PK) profile) with time-matched, placebo-corrected, baseline-adjusted difference in QTcF interval (delta delta QTcF); and the PK and safety profiles of the new zoliflodacin formulation. Each subject will receive one dose of each of four treatments: zoliflodacin 2 g orally, zoliflodacin 4 g orally, placebo for zoliflodacin 4 g orally, and moxifloxacin 400 mg orally. The study will last approximately 12 weeks with a subject participation duration of up to 55 days. The primary hypothesis to be tested is that following administration of zoliflodacin 2 g and 4 g, the upper bound of the one-sided 95% confidence interval (CI) of treatment effect on delta delta QTcF is > / = 10 msec for at least one of the ECG assessments, against the alternative hypothesis that all mean effects are < 10 msec. The primary objective is to evaluate the effect of zoliflodacin on the corrected QT interval of the ECG using Fridericia's formula (QTcF).

DETAILED DESCRIPTION:
The Phase I Thorough QT/QTc (TQT) study will be performed in a single center, the Vince & Associates Clinical Research, Inc., clinical trials unit (CTU), according to a randomized, double-blinded (except for the use of moxifloxacin), placebo-controlled, four-period, four-treatment, crossover design balanced with respect to first-order carryover effect in 72 healthy male or female subjects, aged 18 to 45 years inclusive, to evaluate the effect of zoliflodacin on the corrected QT interval of the electrocardiogram (ECG) using Fridericia's Formula (QTcF) and other ECG parameters; the correlation of the drug concentrations (and pharmacokinetic (PK) profile) with time-matched, placebo-corrected, baseline-adjusted difference in QTcF interval (delta delta QTcF); and the PK and safety profiles of the new zoliflodacin formulation. Each subject will receive one dose of each of four treatments: zoliflodacin 2 g orally, zoliflodacin 4 g orally, placebo for zoliflodacin 4 g orally, and moxifloxacin 400 mg orally. The study will last approximately 12 weeks with a subject participation duration of up to 55 days. The primary hypothesis to be tested is that following administration of zoliflodacin 2 g and 4 g, the upper bound of the one-sided 95% confidence interval (CI) of treatment effect on delta delta QTcF is > / = 10 msec for at least one of the ECG assessments, against the alternative hypothesis that all mean effects are < 10 msec. The primary objective is to evaluate the effect of zoliflodacin on the corrected QT interval of the ECG using Fridericia's formula (QTcF). The secondary objectives are: 1) to evaluate the effects of zoliflodacin on other ECG parameters (PR, QRS, and RR intervals, and heart rate (HR)); 2) to evaluate the sensitivity of QTcF measurement using moxifloxacin; 3) to evaluate the effect of zoliflodacin on T-wave morphology; 4) to evaluate the PK of 2 g and 4 g oral zoliflodacin under fasting state; 5) to evaluate the relationship between zoliflodacin PK and time-matched QTcF pharmacodynamics (PD); 6) to evaluate the safety and tolerability of 2 g and 4 g oral zoliflodacin.

ELIGIBILITY:
Inclusion Criteria:

All must be answered YES for the subject to be eligible for study participation:

1. Informed consent form (ICF) understood and signed before initiating any study procedures
2. Healthy male or female, as assessed by authorized site clinician (listed on FDA Form 1572)
3. Willingness to comply with and be available for all protocol procedures, including inpatient confinement for 3 days in each dosing period and follow-up for the duration of the trial
4. Aged 18 to 45 years inclusive on the day of first dosing
5. Body Mass Index (BMI) > / = 18.5 and < / = to 30 kg per m^2 and weight > / = 50 kg (110 lbs.) and < / = 100 kg (220 lbs.)
6. In all female subjects, whether of childbearing potential or post-menopausal by medical history (MH), a negative serum pregnancy test at Screening Visit and on Day -1 of each dosing period

   -Note: A woman is considered of childbearing potential unless post-menopausal (> / = 1 year without menses without other known or suspected cause and with a FSH level in the menopausal range), or surgically sterilized (hysterectomy, salpingectomy, oophorectomy, or tubal ligation/occlusion).
7. If female, not pregnant, not breast feeding, and not planning to become pregnant during the trial and for 30 days after Final Visit
8. Females of childbearing potential and males agree to use acceptable contraception for the duration of the trial and for 30 days (females) or 90 days (males) after Final Visit

   -Note: A highly effective method of birth control is defined as one with a low failure rate (i.e., less than 1 percent per year) according to CDC criteria. These include progestin implants, intrauterine devices (IUDs), surgical (hysterectomy, salpingectomy, oophorectomy, or tubal ligation/occlusion; vasectomy), or abstinence. Use of methods with higher failure rate (such as progestin injectables, combined oral hormonal contraceptives, condoms, and diaphragms) will not be acceptable when used alone, but they could be considered if used in combination with another method (e.g., a female using combined oral contraceptives if her male partner is sterile, or if she and her non-sterile male partner use a double-barrier method), after consultation with the DMID Medical Officer.
9. Male subjects agree to refrain from sperm donation for the duration of the trial and for 90 days after Final Visit
10. Laboratory tests are in the normal reference range with acceptable exceptions
11. Vital signs (VS) are within the acceptable range
12. Has adequate venous access for blood collection
13. Urine drug screen is negative for tested substances
14. Urine alcohol test is negative
15. Willing to abstain from alcohol consumption for 2 days before Day -1 of Period 1 and for the duration of the trial

Exclusion Criteria:

All must be answered NO for the subject to be eligible for study participation:

1. History of acute or chronic cardiovascular disease or surgery

* Note: Conditions include: congestive heart failure; coronary artery disease (myocardial infarction, unstable angina); cerebrovascular disease (cerebrovascular accident or stroke or transient ischemic attack (TIA); chronic hypertension; or coronary revascularization surgery (coronary artery bypass grafting or percutaneous transluminal coronary angioplasty) 2. History of cardiac arrhythmia or syncope related to cardiac arrhythmia or unexplained, or use of a cardiac pacemaker
* Note: Conditions include: atrial fibrillation, atrial flutter, or non-sustained or sustained ventricular tachycardia; use of a cardiac pacemaker; personal or family history of LQTS; or family history of sudden death 3. History of any other chronic medical or surgical condition that would interfere with the accurate assessment of the trial's objectives or increase the subject's risk profile
* Note: Chronic medical conditions include: diabetes mellitus; asthma requiring use of medication in the year before screening; autoimmune disorder such as lupus erythematosus, Wegener's, rheumatoid arthritis, thyroid disease; malignancy except low-grade (squamous and basal cell) skin cancer thought to be cured; chronic renal, hepatic, pulmonary, or endocrine disease, myopathy, or neuropathy; gastrointestinal surgery including weight loss surgery or biliary surgery 4. Major surgical interventions are not permitted within 4 weeks of first dosing and during the trial. Minor surgical interventions are not allowed within 2 weeks of first dosing and during the trial 5. History of hypersensitivity or severe allergic reaction of any type to medications, bee stings, food, or environmental factors
* Note: Severe allergic reaction is defined as any of the following: anaphylaxis, urticaria, or angioedema 6. Active allergic symptoms to seasonal and animal allergens that are moderate to severe, affect daily activity, and require continuous treatment 7. A marked baseline prolongation of ECG intervals, or HR less than 45 bpm or greater than 100 bpm on ECG measurements
* Note: The following are considered prolonged ECG intervals: QTc/QTcF > 449 msec in males and females; PR > 209 msec; and QRS > 110 msec 8. Clinically significant abnormal ECG results
* Note: Clinically significant abnormal ECG results include: complete left or right bundle branch block; other ventricular conduction block; 2nd degree or 3rd degree atrioventricular (AV) block; sustained atrial or ventricular arrhythmia; two premature ventricular contractions in a row; pattern of ST elevation felt consistent with cardiac ischemia; evidence of a previous myocardial infarction (MI), left ventricular hypertrophy (LVH), or more than minor non-specific ST-T wave changes; any characteristics that would make QT assessment unreliable, including flat T waves; or any condition deemed clinically significant by a study investigator 9. Abnormal renal function
* Note: Normal renal function is defined as normal creatinine and normal estimated glomerular filtration rate (eGFR) [i.e., > 80.0 mL/min] values according to Cockroft-Gault 10. Positive serology results for HIV, HBsAg, or HCV 11. Febrile illness with temperature > / = 38.0 degrees Celsius for < 7 days before dosing in each treatment period 12. Donated whole blood or blood products within 60 days before first dosing, or plans to donate or receive before Final Visit (Day 8 + / - 2 after last dose in dosing period 4)
* Note: Blood products include RBCs, white blood cells (WBCs), platelets, and plasma 13. Known allergic reactions to fluoroquinolones or to components present in the formulation or processing of zoliflodacin and moxifloxacin 14. Treatment with another investigational product within 30 days of first dosing or 5 half-lives or twice the duration of the biological effect of the study drug (whichever is longer)
* Note: Investigational products include a drug, vaccine, biologic, device, or blood product 15. Active drug or alcohol binge consumption, abuse, or dependence within 12 months before Screening Visit that, in the opinion of the investigator, would interfere with adherence to study requirements 16. Use of any prescription medication within 30 days before first dosing or planned use during the trial except as noted below and approved by the designated study clinician
* Note 1: Prohibited medications include moderate or strong CYP3A4 inducers and other drugs with known risk for QT prolongation and TdP; antibiotics; injectable or oral antidiabetic drugs; anti-lipid drugs; immunosuppressive agents; immune modulators; oral corticosteroids; anti-neoplastic agents; any vaccine (licensed or investigational) except licensed influenza vaccine during the flu season, which is allowed up to 7 days before first dosing or 7 days after last dosing
* Note 2: Allowed medications include: oral contraceptives; H1 antihistamines; all medications approved for control of intraocular pressure including topical ophthalmic non-selective beta-blockers, such as betaxolol, carteolol, levobunolol, metipranolol, and timolol; topical/ intranasal corticosteroids; nonsteroidal anti-inflammatory drugs (NSAIDS); licensed influenza vaccine during the flu season, 7 days before first dosing or 7 days after last dosing 17. Use of non-prescription medications, vitamins, herbs, or nutritional supplements within 15 days before first dosing or planned use during the trial unless approved by the study clinician
* Note 1: Intake of nutritional supplements, juice, and herbal preparations or other foods or beverages that may affect the various drug-metabolizing enzymes and transporters (e.g., grapefruit, grapefruit juice, grapefruit-containing beverages, apple or orange juice, vegetables from the mustard green family [e.g., kale, broccoli, watercress, collard greens, kohlrabi, Brussels sprouts, mustard], and charbroiled meats) within 7 days before dosing
* Note 2: Exceptions: St. John's wart is not allowed within 30 days of dosing; vitamins and over-the-counter (OTC) medications taken for a brief period (less than 48 h) for the treatment of common symptoms (such as headache, indigestion, muscle pain) may be allowed as approved by the designated study clinician 18. Intake of caffeinated beverages or food within 72 h before first dosing or a history of high caffeine consumption (e.g., in the last 4 months drinking > 5 cups of coffee/day) 19. Smoking or use of tobacco or nicotine-containing products within 30 days before first dosing 20. Engagement in strenuous exercise within 15 days before first dosing (e.g., marathon running, long-distance cycling, weight lifting) and during the trial 21. Any specific behavioral or clinical condition that, in the judgment of the investigator, precludes participation because it could affect compliance with study procedures or subject safety 22. Plans to enroll or is already enrolled in another clinical trial that could interfere with safety assessment of the study drug at any time during the trial
* Note: Includes trials that have a study intervention such as a drug, biologic, or device 23. Is a CTU employee or staff member who is paid entirely or partially by the Office of Clinical Research Resources (OCRR)/NIAID contract for the DMID-funded trial
* Note: CTU employees or staff include the PIs, sub-investigators, or staff who are supervised by the PI or sub-investigators

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2018-09-25 (Actual); Primary Completion 2019-01-02 (Actual); Study Completion 2019-01-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Vince and Associates Clinical Research, Overland Park, Kansas, United States

REFERENCES:
- [Derived] Newman LM, Kankam M, Nakamura A, Conrad T, Mueller J, O'Donnell J, Osborn BL, Gu K, Saviolakis GA. Thorough QT Study To Evaluate the Effect of Zoliflodacin, a Novel Therapeutic for Gonorrhea, on Cardiac Repolarization in Healthy Adults. Antimicrob Agents Chemother. 2021 Nov 17;65(12):e0129221. doi: 10.1128/AAC.01292-21. Epub 2021 Oct 4. PMID 34606332

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was performed at a commercial phase 1 unit. Recruitment opened on September 4, 2018 and all 72 participants were consented and screened for meeting eligibility criteria prior to enrollment and dosing. Enrollment was completed on December 04, 2018.
Groups:
- 2g Zoliflodacin, 4g Zoliflodacin, Placebo, 400mg Moxifloxacin: Treatment ABCD: 2 g of zoliflodacin administered orally on Day 1, then an 8 day wash out 4 g of zoliflodacin was taken, then another 8 day wash out placebo was taken and then after the final 8 day wash out 400mg of moxifloxacin was taken.
  AZD0914: Spiropyrimidinetrione antibacterial drug, powder (zoliflodacin) was reconstituted in 60 mL of water and dosed orally following an overnight fast, after which approximately 60 mL of water was added to the cup and consumed by the subject.
  Placebo: Composed of 4g of the same excipients found in zoliflodacin. Powder was reconstituted in 60 mL of water and dosed orally. After the cup containing 60 mL of placebo was taken, approximately 60 mL of water was consumed by the subject to chase the initial dose.
  Moxifloxacin: Broad-spectrum 8-methoxy fluoroquinolone. A single, commercially-available, film-coated, 400-mg tablet of moxifloxacin hydrochloride was administered orally with 120 mL of water.
- 2g Zoliflodacin, Placebo, 400mg Moxifloxacin, 4g Zoliflodacin: Treatment ACDB: 2 g of zoliflodacin administered orally on Day 1, then an 8 day wash out placebo was taken, then another 8 day wash out, 400 mg moxifloxacin was taken and then after the final 8 day wash out 4 g of zoliflodacin was taken.
  AZD0914: Spiropyrimidinetrione antibacterial drug, powder (zoliflodacin) was reconstituted in 60 mL of water and dosed orally following an overnight fast, after which approximately 60 mL of water was added to the cup and consumed by the subject.
  Placebo: Composed of 4g of the same excipients found in zoliflodacin. Powder was reconstituted in 60 mL of water and dosed orally. After the cup containing 60 mL of placebo was taken, approximately 60 mL of water was consumed by the subject to chase the initial dose.
  Moxifloxacin: Broad-spectrum 8-methoxy fluoroquinolone. A single, commercially-available, film-coated, 400-mg tablet of moxifloxacin hydrochloride was administered orally with 120 mL of water.
- 2g Zoliflodacin, 400mg Moxifloxacin, 4g Zoliflodacin, Placebo: Treatment ADBC: 2 g of zoliflodacin administered orally on Day 1, then an 8 day wash out 400mg of moxifloxacin was taken, then another 8 day wash out 4g of zoliflodacin was taken and then after the final 8 day wash out placebo was taken.
  AZD0914: Spiropyrimidinetrione antibacterial drug, powder (zoliflodacin) was reconstituted in 60 mL of water and dosed orally following an overnight fast, after which approximately 60 mL of water was added to the cup and consumed by the subject.
  Placebo: Composed of 4g of the same excipients found in zoliflodacin. Powder was reconstituted in 60 mL of water and dosed orally. After the cup containing 60 mL of placebo was taken, approximately 60 mL of water was consumed by the subject to chase the initial dose.
  Moxifloxacin: Broad-spectrum 8-methoxy fluoroquinolone. A single, commercially-available, film-coated, 400-mg tablet of moxifloxacin hydrochloride was administered orally with 120 mL of water.
- 4g Zoliflodacin, 2g Zoliflodacin, 400mg Moxifloxacin, Placebo: Treatment BADC: 4 g of zoliflodacin administered orally on Day 1, then an 8 day wash out 2 g of zoliflodacin was taken, then another 8 day wash out 400mg of moxifloxacin was taken and then after the final 8 day wash out placebo was taken.
  AZD0914: Spiropyrimidinetrione antibacterial drug, powder (zoliflodacin) was reconstituted in 60 mL of water and dosed orally following an overnight fast, after which approximately 60 mL of water was added to the cup and consumed by the subject.
  Placebo: Composed of 4g of the same excipients found in zoliflodacin. Powder was reconstituted in 60 mL of water and dosed orally. After the cup containing 60 mL of placebo was taken, approximately 60 mL of water was consumed by the subject to chase the initial dose.
  Moxifloxacin: Broad-spectrum 8-methoxy fluoroquinolone. A single, commercially-available, film-coated, 400-mg tablet of moxifloxacin hydrochloride was administered orally with 120 mL of water.
- 4g Zoliflodacin, 400mg Moxifloxacin, Placebo, 2g Zoliflodacin,: Treatment BDCA: 4 g of zoliflodacin administered orally on Day 1, then an 8 day wash out 400mg of moxifloxacin was taken, then another 8 day wash out placebo was taken and then after the final 8 day wash out 2 g of zoliflodacin was taken.
  AZD0914: Spiropyrimidinetrione antibacterial drug, powder (zoliflodacin) was reconstituted in 60 mL of water and dosed orally following an overnight fast, after which approximately 60 mL of water was added to the cup and consumed by the subject.
  Placebo: Composed of 4g of the same excipients found in zoliflodacin. Powder was reconstituted in 60 mL of water and dosed orally. After the cup containing 60 mL of placebo was taken, approximately 60 mL of water was consumed by the subject to chase the initial dose.
  Moxifloxacin: Broad-spectrum 8-methoxy fluoroquinolone. A single, commercially-available, film-coated, 400-mg tablet of moxifloxacin hydrochloride was administered orally with 120 mL of water.
- 4g Zoliflodacin, Placebo, 2g Zoliflodacin, 400mg Moxifloxacin: Treatment BCAD: 4 g of zoliflodacin administered orally on Day 1, then an 8 day wash out placebo was taken, then another 8 day wash out 2 g of zoliflodacin was taken and then after the final 8 day wash out 400mg of moxifloxacin was taken.
  AZD0914: Spiropyrimidinetrione antibacterial drug, powder (zoliflodacin) was reconstituted in 60 mL of water and dosed orally following an overnight fast, after which approximately 60 mL of water was added to the cup and consumed by the subject.
  Placebo: Composed of 4g of the same excipients found in zoliflodacin. Powder was reconstituted in 60 mL of water and dosed orally. After the cup containing 60 mL of placebo was taken, approximately 60 mL of water was consumed by the subject to chase the initial dose.
  Moxifloxacin: Broad-spectrum 8-methoxy fluoroquinolone. A single, commercially-available, film-coated, 400-mg tablet of moxifloxacin hydrochloride was administered orally with 120 mL of water.
- Placebo, 400mg Moxifloxacin, 2g Zoliflodacin, 4g Zoliflodacin,: Treatment CDAB: Placebo administered orally on Day 1, then an 8 day wash out 400mg of moxifloxacin was taken, then another 8 day wash out 2 g of zoliflodacin was taken and then after the final 8 day wash out 4 g of zoliflodacin was taken.
  AZD0914: Spiropyrimidinetrione antibacterial drug, powder (zoliflodacin) was reconstituted in 60 mL of water and dosed orally following an overnight fast, after which approximately 60 mL of water was added to the cup and consumed by the subject.
  Placebo: Composed of 4g of the same excipients found in zoliflodacin. Powder was reconstituted in 60 mL of water and dosed orally. After the cup containing 60 mL of placebo was taken, approximately 60 mL of water was consumed by the subject to chase the initial dose.
  Moxifloxacin: Broad-spectrum 8-methoxy fluoroquinolone. A single, commercially-available, film-coated, 400-mg tablet of moxifloxacin hydrochloride was administered orally with 120 mL of water.
- Placebo, 2g Zoliflodacin, 4g Zoliflodacin, 400mg Moxifloxacin: Treatment CABD: Placebo administered orally on Day 1, then an 8 day wash out 2 g of zoliflodacin was taken, then another 8 day wash out 4 g of zoliflodacin was taken and then after the final 8 day wash out 400mg of moxifloxacin was taken.
  AZD0914: Spiropyrimidinetrione antibacterial drug, powder (zoliflodacin) was reconstituted in 60 mL of water and dosed orally following an overnight fast, after which approximately 60 mL of water was added to the cup and consumed by the subject.
  Placebo: Composed of 4g of the same excipients found in zoliflodacin. Powder was reconstituted in 60 mL of water and dosed orally. After the cup containing 60 mL of placebo was taken, approximately 60 mL of water was consumed by the subject to chase the initial dose.
  Moxifloxacin: Broad-spectrum 8-methoxy fluoroquinolone. A single, commercially-available, film-coated, 400-mg tablet of moxifloxacin hydrochloride was administered orally with 120 mL of water.
- Placebo, 4g Zoliflodacin, 400mg Moxifloxacin, 2g Zoliflodacin: Treatment CBDA: Placebo administered orally on Day 1, then an 8 day wash out 4 g of zoliflodacin was taken, then another 8 day wash out 400mg of moxifloxacin was taken and then after the final 8 day wash out 2 g of zoliflodacin was taken.
  AZD0914: Spiropyrimidinetrione antibacterial drug, powder (zoliflodacin) was reconstituted in 60 mL of water and dosed orally following an overnight fast, after which approximately 60 mL of water was added to the cup and consumed by the subject.
  Placebo: Composed of 4g of the same excipients found in zoliflodacin. Powder was reconstituted in 60 mL of water and dosed orally. After the cup containing 60 mL of placebo was taken, approximately 60 mL of water was consumed by the subject to chase the initial dose.
  Moxifloxacin: Broad-spectrum 8-methoxy fluoroquinolone. A single, commercially-available, film-coated, 400-mg tablet of moxifloxacin hydrochloride was administered orally with 120 mL of water.
- 400mg Moxifloxacin, Placebo, 4g Zoliflodacin, 2g Zoliflodacin: Treatment DCBA: 400mg of moxifloxacin was administered orally on Day 1, then an 8 day wash out placebo was taken, then another 8 day wash out 4 g of zoliflodacin was taken and then after the final 8 day wash out 2 g of zoliflodacin was taken.
  AZD0914: Spiropyrimidinetrione antibacterial drug, powder (zoliflodacin) was reconstituted in 60 mL of water and dosed orally following an overnight fast, after which approximately 60 mL of water was added to the cup and consumed by the subject.
  Placebo: Composed of 4g of the same excipients found in zoliflodacin. Powder was reconstituted in 60 mL of water and dosed orally. After the cup containing 60 mL of placebo was taken, approximately 60 mL of water was consumed by the subject to chase the initial dose.
  Moxifloxacin: Broad-spectrum 8-methoxy fluoroquinolone. A single, commercially-available, film-coated, 400-mg tablet of moxifloxacin hydrochloride was administered orally with 120 mL of water.
- 400mg Moxifloxacin, 4g Zoliflodacin, 2g Zoliflodacin, Placebo: Treatment DBAC: 400mg of moxifloxacin was administered orally on Day 1, then an 8 day wash out 4 g of zoliflodacin was taken, then another 8 day wash out 2 g of zoliflodacin was taken and then after the final 8 day wash out placebo was taken.
  AZD0914: Spiropyrimidinetrione antibacterial drug, powder (zoliflodacin) was reconstituted in 60 mL of water and dosed orally following an overnight fast, after which approximately 60 mL of water was added to the cup and consumed by the subject.
  Placebo: Composed of 4g of the same excipients found in zoliflodacin. Powder was reconstituted in 60 mL of water and dosed orally. After the cup containing 60 mL of placebo was taken, approximately 60 mL of water was consumed by the subject to chase the initial dose.
  Moxifloxacin: Broad-spectrum 8-methoxy fluoroquinolone. A single, commercially-available, film-coated, 400-mg tablet of moxifloxacin hydrochloride was administered orally with 120 mL of water.
- 400mg Moxifloxacin, 2g Zoliflodacin, Placebo, 4g Zoliflodacin: Treatment DACB: 400mg of moxifloxacin was administered orally on Day 1, then an 8 day wash out 2 g of zoliflodacin was taken, then another 8 day wash out placebo was taken and then after the final 8 day wash out 4 g of zoliflodacin was taken.
  AZD0914: Spiropyrimidinetrione antibacterial drug, powder (zoliflodacin) was reconstituted in 60 mL of water and dosed orally following an overnight fast, after which approximately 60 mL of water was added to the cup and consumed by the subject.
  Placebo: Composed of 4g of the same excipients found in zoliflodacin. Powder was reconstituted in 60 mL of water and dosed orally. After the cup containing 60 mL of placebo was taken, approximately 60 mL of water was consumed by the subject to chase the initial dose.
  Moxifloxacin: Broad-spectrum 8-methoxy fluoroquinolone. A single, commercially-available, film-coated, 400-mg tablet of moxifloxacin hydrochloride was administered orally with 120 mL of water.
Period: First Treatment
Arm/Group | 2g Zoliflodacin, 4g Zoliflodacin, Placebo, 400mg Moxifloxacin | 2g Zoliflodacin, Placebo, 400mg Moxifloxacin, 4g Zoliflodacin | 2g Zoliflodacin, 400mg Moxifloxacin, 4g Zoliflodacin, Placebo | 4g Zoliflodacin, 2g Zoliflodacin, 400mg Moxifloxacin, Placebo | 4g Zoliflodacin, 400mg Moxifloxacin, Placebo, 2g Zoliflodacin, | 4g Zoliflodacin, Placebo, 2g Zoliflodacin, 400mg Moxifloxacin | Placebo, 400mg Moxifloxacin, 2g Zoliflodacin, 4g Zoliflodacin, | Placebo, 2g Zoliflodacin, 4g Zoliflodacin, 400mg Moxifloxacin | Placebo, 4g Zoliflodacin, 400mg Moxifloxacin, 2g Zoliflodacin | 400mg Moxifloxacin, Placebo, 4g Zoliflodacin, 2g Zoliflodacin | 400mg Moxifloxacin, 4g Zoliflodacin, 2g Zoliflodacin, Placebo | 400mg Moxifloxacin, 2g Zoliflodacin, Placebo, 4g Zoliflodacin
Started | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
Received Treatment | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
Completed | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Second Treatment
Arm/Group | 2g Zoliflodacin, 4g Zoliflodacin, Placebo, 400mg Moxifloxacin | 2g Zoliflodacin, Placebo, 400mg Moxifloxacin, 4g Zoliflodacin | 2g Zoliflodacin, 400mg Moxifloxacin, 4g Zoliflodacin, Placebo | 4g Zoliflodacin, 2g Zoliflodacin, 400mg Moxifloxacin, Placebo | 4g Zoliflodacin, 400mg Moxifloxacin, Placebo, 2g Zoliflodacin, | 4g Zoliflodacin, Placebo, 2g Zoliflodacin, 400mg Moxifloxacin | Placebo, 400mg Moxifloxacin, 2g Zoliflodacin, 4g Zoliflodacin, | Placebo, 2g Zoliflodacin, 4g Zoliflodacin, 400mg Moxifloxacin | Placebo, 4g Zoliflodacin, 400mg Moxifloxacin, 2g Zoliflodacin | 400mg Moxifloxacin, Placebo, 4g Zoliflodacin, 2g Zoliflodacin | 400mg Moxifloxacin, 4g Zoliflodacin, 2g Zoliflodacin, Placebo | 400mg Moxifloxacin, 2g Zoliflodacin, Placebo, 4g Zoliflodacin
Started | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
Received Treatment | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
Completed | 6 | 6 | 5 | 6 | 5 | 6 | 6 | 6 | 6 | 6 | 6 | 6
Not Completed | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Third Treatment
Arm/Group | 2g Zoliflodacin, 4g Zoliflodacin, Placebo, 400mg Moxifloxacin | 2g Zoliflodacin, Placebo, 400mg Moxifloxacin, 4g Zoliflodacin | 2g Zoliflodacin, 400mg Moxifloxacin, 4g Zoliflodacin, Placebo | 4g Zoliflodacin, 2g Zoliflodacin, 400mg Moxifloxacin, Placebo | 4g Zoliflodacin, 400mg Moxifloxacin, Placebo, 2g Zoliflodacin, | 4g Zoliflodacin, Placebo, 2g Zoliflodacin, 400mg Moxifloxacin | Placebo, 400mg Moxifloxacin, 2g Zoliflodacin, 4g Zoliflodacin, | Placebo, 2g Zoliflodacin, 4g Zoliflodacin, 400mg Moxifloxacin | Placebo, 4g Zoliflodacin, 400mg Moxifloxacin, 2g Zoliflodacin | 400mg Moxifloxacin, Placebo, 4g Zoliflodacin, 2g Zoliflodacin | 400mg Moxifloxacin, 4g Zoliflodacin, 2g Zoliflodacin, Placebo | 400mg Moxifloxacin, 2g Zoliflodacin, Placebo, 4g Zoliflodacin
Started | 6 | 6 | 5 | 6 | 5 | 6 | 6 | 6 | 6 | 6 | 6 | 6
Received Treatment | 6 | 6 | 5 | 6 | 5 | 6 | 5 | 6 | 6 | 6 | 6 | 6
Completed | 6 | 6 | 5 | 6 | 4 | 6 | 5 | 6 | 6 | 6 | 6 | 4
Not Completed | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 2
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Period: Fourth Treatment
Arm/Group | 2g Zoliflodacin, 4g Zoliflodacin, Placebo, 400mg Moxifloxacin | 2g Zoliflodacin, Placebo, 400mg Moxifloxacin, 4g Zoliflodacin | 2g Zoliflodacin, 400mg Moxifloxacin, 4g Zoliflodacin, Placebo | 4g Zoliflodacin, 2g Zoliflodacin, 400mg Moxifloxacin, Placebo | 4g Zoliflodacin, 400mg Moxifloxacin, Placebo, 2g Zoliflodacin, | 4g Zoliflodacin, Placebo, 2g Zoliflodacin, 400mg Moxifloxacin | Placebo, 400mg Moxifloxacin, 2g Zoliflodacin, 4g Zoliflodacin, | Placebo, 2g Zoliflodacin, 4g Zoliflodacin, 400mg Moxifloxacin | Placebo, 4g Zoliflodacin, 400mg Moxifloxacin, 2g Zoliflodacin | 400mg Moxifloxacin, Placebo, 4g Zoliflodacin, 2g Zoliflodacin | 400mg Moxifloxacin, 4g Zoliflodacin, 2g Zoliflodacin, Placebo | 400mg Moxifloxacin, 2g Zoliflodacin, Placebo, 4g Zoliflodacin
Started | 6 | 6 | 5 | 6 | 4 | 6 | 5 | 6 | 6 | 6 | 6 | 4
Received Treatment | 5 | 6 | 5 | 6 | 4 | 6 | 4 | 6 | 6 | 6 | 6 | 4
Completed | 5 | 6 | 5 | 6 | 3 | 6 | 4 | 6 | 6 | 6 | 6 | 4
Not Completed | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- 2g Zoliflodacin, 4g Zoliflodacin, Placebo, 400mg Moxifloxacin: Treatment ABCD: 2 g of zoliflodacin administered orally on Day 1, then an 8 day wash out 4 g of zoliflodacin was taken, then another 8 day wash out placebo was taken and then after the final 8 day wash out 400mg of moxifloxacin was taken.
  AZD0914: Spiropyrimidinetrione antibacterial drug, Powder was reconstituted in 60 mL of water and dosed orally after an overnight fast. After the cup containing 60 mL of zoliflodacin was taken, approximately 60 mL of water was added and consumed by the subject to chase the initial dose.
  Placebo: Composed of 4g of the same excipients found in zoliflodacin. Powder was reconstituted in 60 mL of water and dosed orally. After the cup containing 60 mL of placebo was taken, approximately 60 mL of water was consumed by the subject to chase the initial dose.
  Moxifloxacin: Broad-spectrum 8-methoxy fluoroquinolone. A single, commercially-available, film-coated, 400-mg tablet of moxifloxacin hydrochloride was administered orally with 120 mL of water.
- 2g Zoliflodacin, Placebo, 400mg Moxifloxacin, 4g Zoliflodacin: Treatment ACDB: 2 g of zoliflodacin administered orally on Day 1, then an 8 day wash out placebo was taken, then another 8 day wash out, 400 mg moxifloxacin was taken and then after the final 8 day wash out 4 g of zoliflodacin was taken.
  AZD0914: Spiropyrimidinetrione antibacterial drug, Powder was reconstituted in 60 mL of water and dosed orally after an overnight fast. After the cup containing 60 mL of zoliflodacin was taken, approximately 60 mL of water was added and consumed by the subject to chase the initial dose.
  Placebo: Composed of 4g of the same excipients found in zoliflodacin. Powder was reconstituted in 60 mL of water and dosed orally. After the cup containing 60 mL of placebo was taken, approximately 60 mL of water was consumed by the subject to chase the initial dose.
  Moxifloxacin: Broad-spectrum 8-methoxy fluoroquinolone. A single, commercially-available, film-coated, 400-mg tablet of moxifloxacin hydrochloride was administered orally with 120 mL of water..
- 2g Zoliflodacin, 400mg Moxifloxacin, 4g Zoliflodacin, Placebo: Treatment ADBC: 2 g of zoliflodacin administered orally on Day 1, then an 8 day wash out 400mg of moxifloxacin was taken, then another 8 day wash out 4g of zoliflodacin was taken and then after the final 8 day wash out placebo was taken.
  AZD0914: Spiropyrimidinetrione antibacterial drug, Powder was reconstituted in 60 mL of water and dosed orally after an overnight fast. After the cup containing 60 mL of zoliflodacin was taken, approximately 60 mL of water was added and consumed by the subject to chase the initial dose.
  Placebo: Composed of 4g of the same excipients found in zoliflodacin. Powder was reconstituted in 60 mL of water and dosed orally. After the cup containing 60 mL of placebo was taken, approximately 60 mL of water was consumed by the subject to chase the initial dose.
  Moxifloxacin: Broad-spectrum 8-methoxy fluoroquinolone. A single, commercially-available, film-coated, 400-mg tablet of moxifloxacin hydrochloride was administered orally with 120 mL of water.
- 4g Zoliflodacin, 2g Zoliflodacin, 400mg Moxifloxacin, Placebo: Treatment BADC: 4 g of zoliflodacin administered orally on Day 1, then an 8 day wash out2 g of zoliflodacin was taken, then another 8 day wash out 400mg of moxifloxacin was taken and then after the final 8 day wash out placebo was taken.
  AZD0914: Spiropyrimidinetrione antibacterial drug, Powder was reconstituted in 60 mL of water and dosed orally after an overnight fast. After the cup containing 60 mL of zoliflodacin was taken, approximately 60 mL of water was added and consumed by the subject to chase the initial dose.
  Placebo: Composed of 4g of the same excipients found in zoliflodacin. Powder was reconstituted in 60 mL of water and dosed orally. After the cup containing 60 mL of placebo was taken, approximately 60 mL of water was consumed by the subject to chase the initial dose.
  Moxifloxacin: Broad-spectrum 8-methoxy fluoroquinolone. A single, commercially-available, film-coated, 400-mg tablet of moxifloxacin hydrochloride was administered orally with 120 mL of water.
- 4g Zoliflodacin, 400mg Moxifloxacin, Placebo, 2g Zoliflodacin,: Treatment BDCA: 4 g of zoliflodacin administered orally on Day 1, then an 8 day wash out 400mg of moxifloxacin was taken, then another 8 day wash out placebo was taken and then after the final 8 day wash out 2 g of zoliflodacin was taken.
  AZD0914: Spiropyrimidinetrione antibacterial drug, Powder was reconstituted in 60 mL of water and dosed orally after an overnight fast. After the cup containing 60 mL of zoliflodacin was taken, approximately 60 mL of water was added and consumed by the subject to chase the initial dose.
  Placebo: Composed of 4g of the same excipients found in zoliflodacin. Powder was reconstituted in 60 mL of water and dosed orally. After the cup containing 60 mL of placebo was taken, approximately 60 mL of water was consumed by the subject to chase the initial dose.
  Moxifloxacin: Broad-spectrum 8-methoxy fluoroquinolone. A single, commercially-available, film-coated, 400-mg tablet of moxifloxacin hydrochloride was administered orally with 120 mL of water.
- 4g Zoliflodacin, Placebo, 2g Zoliflodacin, 400mg Moxifloxacin: Treatment BCAD: 4 g of zoliflodacin administered orally on Day 1, then an 8 day wash out placebo was taken, then another 8 day wash out 2 g of zoliflodacin was taken and then after the final 8 day wash out 400mg of moxifloxacin was taken.
  AZD0914: Spiropyrimidinetrione antibacterial drug, Powder was reconstituted in 60 mL of water and dosed orally after an overnight fast. After the cup containing 60 mL of zoliflodacin was taken, approximately 60 mL of water was added and consumed by the subject to chase the initial dose.
  Placebo: Composed of 4g of the same excipients found in zoliflodacin. Powder was reconstituted in 60 mL of water and dosed orally. After the cup containing 60 mL of placebo was taken, approximately 60 mL of water was consumed by the subject to chase the initial dose.
  Moxifloxacin: Broad-spectrum 8-methoxy fluoroquinolone. A single, commercially-available, film-coated, 400-mg tablet of moxifloxacin hydrochloride was administered orally with 120 mL of water.
- Placebo, 400mg Moxifloxacin, 2g Zoliflodacin, 4g Zoliflodacin,: Treatment CDAB: Placebo administered orally on Day 1, then an 8 day wash out 400mg of moxifloxacin was taken, then another 8 day wash out 2 g of zoliflodacin was taken and then after the final 8 day wash out4 g of zoliflodacin was taken.
  AZD0914: Spiropyrimidinetrione antibacterial drug, Powder was reconstituted in 60 mL of water and dosed orally after an overnight fast. After the cup containing 60 mL of zoliflodacin was taken, approximately 60 mL of water was added and consumed by the subject to chase the initial dose.
  Placebo: Composed of 4g of the same excipients found in zoliflodacin. Powder was reconstituted in 60 mL of water and dosed orally. After the cup containing 60 mL of placebo was taken, approximately 60 mL of water was consumed by the subject to chase the initial dose.
  Moxifloxacin: Broad-spectrum 8-methoxy fluoroquinolone. A single, commercially-available, film-coated, 400-mg tablet of moxifloxacin hydrochloride was administered orally with 120 mL of water.
- Placebo, 2g Zoliflodacin, 4g Zoliflodacin, 400mg Moxifloxacin: Treatment CABD: Placebo administered orally on Day 1, then an 8 day wash out 2 g of zoliflodacin was taken, then another 8 day wash out 4 g of zoliflodacin was taken and then after the final 8 day wash out 400mg of moxifloxacin was taken.
  AZD0914: Spiropyrimidinetrione antibacterial drug, Powder was reconstituted in 60 mL of water and dosed orally after an overnight fast. After the cup containing 60 mL of zoliflodacin was taken, approximately 60 mL of water was added and consumed by the subject to chase the initial dose.
  Placebo: Composed of 4g of the same excipients found in zoliflodacin. Powder was reconstituted in 60 mL of water and dosed orally. After the cup containing 60 mL of placebo was taken, approximately 60 mL of water was consumed by the subject to chase the initial dose.
  Moxifloxacin: Broad-spectrum 8-methoxy fluoroquinolone. A single, commercially-available, film-coated, 400-mg tablet of moxifloxacin hydrochloride was administered orally with 120 mL of water.
- Placebo, 4g Zoliflodacin, 400mg Moxifloxacin, 2g Zoliflodacin: Treatment CBDA: Placebo administered orally on Day 1, then an 8 day wash out 4 g of zoliflodacin was taken, then another 8 day wash out 400mg of moxifloxacin was taken and then after the final 8 day wash out 2 g of zoliflodacin was taken.
  AZD0914: Spiropyrimidinetrione antibacterial drug, Powder was reconstituted in 60 mL of water and dosed orally after an overnight fast. After the cup containing 60 mL of zoliflodacin was taken, approximately 60 mL of water was added and consumed by the subject to chase the initial dose.
  Placebo: Composed of 4g of the same excipients found in zoliflodacin. Powder was reconstituted in 60 mL of water and dosed orally. After the cup containing 60 mL of placebo was taken, approximately 60 mL of water was consumed by the subject to chase the initial dose.
  Moxifloxacin: Broad-spectrum 8-methoxy fluoroquinolone. A single, commercially-available, film-coated, 400-mg tablet of moxifloxacin hydrochloride was administered orally with 120 mL of water.
- 400mg Moxifloxacin, Placebo, 4g Zoliflodacin, 2g Zoliflodacin: Treatment DCBA: 400mg of moxifloxacin was administered orally on Day 1, then an 8 day wash out placebo was taken, then another 8 day wash out 4 g of zoliflodacin was taken and then after the final 8 day wash out 2 g of zoliflodacin was taken.
  AZD0914: Spiropyrimidinetrione antibacterial drug, Powder was reconstituted in 60 mL of water and dosed orally after an overnight fast. After the cup containing 60 mL of zoliflodacin was taken, approximately 60 mL of water was added and consumed by the subject to chase the initial dose.
  Placebo: Composed of 4g of the same excipients found in zoliflodacin. Powder was reconstituted in 60 mL of water and dosed orally. After the cup containing 60 mL of placebo was taken, approximately 60 mL of water was consumed by the subject to chase the initial dose.
  Moxifloxacin: Broad-spectrum 8-methoxy fluoroquinolone. A single, commercially-available, film-coated, 400-mg tablet of moxifloxacin hydrochloride was administered orally with 120 mL of water.
- 400mg Moxifloxacin, 4g Zoliflodacin, 2g Zoliflodacin, Placebo: Treatment DBAC: 400mg of moxifloxacin was administered orally on Day 1, then an 8 day wash out 4 g of zoliflodacin was taken, then another 8 day wash out 2 g of zoliflodacin was taken and then after the final 8 day wash out placebo was taken.
  AZD0914: Spiropyrimidinetrione antibacterial drug, Powder was reconstituted in 60 mL of water and dosed orally after an overnight fast. After the cup containing 60 mL of zoliflodacin was taken, approximately 60 mL of water was added and consumed by the subject to chase the initial dose.
  Placebo: Composed of 4g of the same excipients found in zoliflodacin. Powder was reconstituted in 60 mL of water and dosed orally. After the cup containing 60 mL of placebo was taken, approximately 60 mL of water was consumed by the subject to chase the initial dose.
  Moxifloxacin: Broad-spectrum 8-methoxy fluoroquinolone. A single, commercially-available, film-coated, 400-mg tablet of moxifloxacin hydrochloride was administered orally with 120 mL of water.
- 400mg Moxifloxacin, 2g Zoliflodacin, Placebo, 4g Zoliflodacin: Treatment DACB: 400mg of moxifloxacin was administered orally on Day 1, then an 8 day wash out 2 g of zoliflodacin was taken, then another 8 day wash out placebo was taken and then after the final 8 day wash out 4 g of zoliflodacin was taken.
  AZD0914: Spiropyrimidinetrione antibacterial drug, Powder was reconstituted in 60 mL of water and dosed orally after an overnight fast. After the cup containing 60 mL of zoliflodacin was taken, approximately 60 mL of water was added and consumed by the subject to chase the initial dose.
  Placebo: Composed of 4g of the same excipients found in zoliflodacin. Powder was reconstituted in 60 mL of water and dosed orally. After the cup containing 60 mL of placebo was taken, approximately 60 mL of water was consumed by the subject to chase the initial dose.
  Moxifloxacin: Broad-spectrum 8-methoxy fluoroquinolone. A single, commercially-available, film-coated, 400-mg tablet of moxifloxacin hydrochloride was administered orally with 120 mL of water.
- Total: Total of all reporting groups
Arm/Group | 2g Zoliflodacin, 4g Zoliflodacin, Placebo, 400mg Moxifloxacin | 2g Zoliflodacin, Placebo, 400mg Moxifloxacin, 4g Zoliflodacin | 2g Zoliflodacin, 400mg Moxifloxacin, 4g Zoliflodacin, Placebo | 4g Zoliflodacin, 2g Zoliflodacin, 400mg Moxifloxacin, Placebo | 4g Zoliflodacin, 400mg Moxifloxacin, Placebo, 2g Zoliflodacin, | 4g Zoliflodacin, Placebo, 2g Zoliflodacin, 400mg Moxifloxacin | Placebo, 400mg Moxifloxacin, 2g Zoliflodacin, 4g Zoliflodacin, | Placebo, 2g Zoliflodacin, 4g Zoliflodacin, 400mg Moxifloxacin | Placebo, 4g Zoliflodacin, 400mg Moxifloxacin, 2g Zoliflodacin | 400mg Moxifloxacin, Placebo, 4g Zoliflodacin, 2g Zoliflodacin | 400mg Moxifloxacin, 4g Zoliflodacin, 2g Zoliflodacin, Placebo | 400mg Moxifloxacin, 2g Zoliflodacin, Placebo, 4g Zoliflodacin | Total
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 72
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 72
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.8 (4.4) | 29.7 (4.7) | 32.5 (4.7) | 36.3 (7.4) | 30.0 (7.3) | 32.5 (8.1) | 31.7 (9.4) | 34.2 (5.5) | 28.7 (4.5) | 30.8 (8.9) | 31.2 (7.1) | 29.0 (6.8) | 31.7 (6.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 2 | 4 | 1 | 4 | 1 | 3 | 1 | 2 | 1 | 2 | 26
  Male | 4 | 3 | 4 | 2 | 5 | 2 | 5 | 3 | 5 | 4 | 5 | 4 | 46
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 0 | 0 | 1 | 2 | 0 | 2 | 0 | 0 | 0 | 3 | 10
  Not Hispanic or Latino | 5 | 5 | 6 | 6 | 5 | 4 | 6 | 4 | 6 | 6 | 6 | 3 | 62
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 3
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 4 | 3 | 4 | 3 | 1 | 2 | 4 | 3 | 2 | 4 | 3 | 2 | 35
  White | 2 | 3 | 2 | 3 | 4 | 4 | 2 | 2 | 4 | 2 | 3 | 3 | 34
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 72
BMI [Mean (Standard Deviation); unit: kg/m^2] | 23.60 (3.20) | 23.98 (2.78) | 24.48 (2.76) | 24.57 (3.28) | 26.10 (2.50) | 25.07 (3.48) | 26.80 (1.58) | 25.67 (2.43) | 23.43 (3.72) | 26.30 (1.68) | 25.35 (3.71) | 25.03 (2.83) | 25.03 (2.87)
Weight [Mean (Standard Deviation); unit: kiliograms] | 71.38 (11.89) | 68.05 (11.16) | 72.65 (14.07) | 70.05 (14.31) | 80.28 (13.93) | 73.63 (14.97) | 80.63 (7.84) | 75.40 (8.74) | 75.57 (17.40) | 78.88 (10.18) | 77.02 (10.28) | 70.85 (14.62) | 74.53 (12.37)

OUTCOME MEASURES:

1. Primary Outcome: The One-sided 95% Confidence Interval (CI) for the Largest Time-matched, Placebo-corrected, Baseline-adjusted Mean QTcF Interval (Delta Delta QTcF) Following Administration of Zoliflodacin
Description: Mean and 90% two-sided confidence intervals (t-intervals) of change from baseline QTcF intervals by time point and treatment. Note that the upper bound of the 90% two-sided confidence interval can also be interpreted as the upper bound of a 95% one-sided confidence interval.
Time Frame: Baseline, 0.5 hour (h), 1 h, 2 h, 3 h, 4 h, 6 h, 8 h, 12 h, and 24 h post-dose after 2 and 4 g zolifloadacin
Population: The analysis population sample size is equal to the number of subjects in the Holter ECG Analysis Population who received a dose of zoliflodacin or a dose of placebo.
Measure: Mean (90% Confidence Interval); unit: milliseconds (msec)
Groups:
- 2 g of Zoliflodacin: 2 g of zoliflodacin administered orally on Day 1 of dosing period.
- 4 g of Zoliflodacin: 4 g of zoliflodacin administered orally on Day 1 of dosing period.
- Placebo: Placebo was administered orally on Day 1 of dosing period.
Arm/Group | 2 g of Zoliflodacin | 4 g of Zoliflodacin | Placebo
Number analyzed (Participants) | 68 | 66 | 69
milliseconds (msec)
  0.5 hour post dose: number analyzed (Participants) | 67 | 65 | 69
  0.5 hour post dose | -3.2 [-4.12 to -2.21] | -1.0 [-2.08 to 0.17] | -2.1 [-2.89 to -1.23]
  1 hour post dose | -1.9 [-2.81 to -1.04] | 0.1 [-1.03 to 1.18] | -2.3 [-3.34 to -1.29]
  2 hour post dose: number analyzed (Participants) | 67 | 66 | 69
  2 hour post dose | -2.3 [-3.43 to -1.25] | 0.1 [-1.25 to 1.47] | -2.2 [-3.30 to -1.19]
  3 hour post dose: number analyzed (Participants) | 67 | 66 | 69
  3 hour post dose | -1.6 [-2.79 to -0.41] | 0.1 [-1.54 to 1.69] | -2.6 [-3.78 to -1.32]
  4 hour post dose: number analyzed (Participants) | 67 | 66 | 69
  4 hour post dose | -2.4 [-3.83 to -0.89] | 0.1 [-1.14 to 1.35] | -3.3 [-4.36 to -2.16]
  6 hour post dose: number analyzed (Participants) | 67 | 66 | 69
  6 hour post dose | -2.0 [-3.50 to -0.50] | -0.7 [-2.37 to 1.07] | -2.3 [-4.55 to -0.06]
  8 hour post dose: number analyzed (Participants) | 67 | 66 | 69
  8 hour post dose | -5.6 [-7.25 to -3.88] | -4.7 [-6.08 to -3.26] | -4.4 [-6.23 to -2.67]
  12 hour post dose: number analyzed (Participants) | 67 | 65 | 69
  12 hour post dose | -2.8 [-4.28 to -1.33] | -0.4 [-2.07 to 1.24] | -2.2 [-4.11 to -0.27]
  24 hour post dose: number analyzed (Participants) | 67 | 64 | 65
  24 hour post dose | -2.9 [-4.17 to -1.53] | -0.3 [-1.49 to 0.93] | -2.2 [-3.69 to -0.77]
Statistical Analysis 1: Comparison: 2 g of Zoliflodacin vs Placebo; Null Hypothesis: Zoliflodacin administered at a 2 g dose causes a prolongation of the QTcF interval 0.5 h post-dose that exceeds the criteria in the ICH Guidance E14 (5 ms). Power Calculation: Enrollment of 72 subjects would provide at least 84% power to conclude a negative effect, given that up to 16 subjects may withdraw early prior to beginning to replace subjects (at least 56 subjects evaluable), and assuming a standard deviation of ΔΔQTcF of 7 msec and an underlying effect of 5 msec; Test type: Non-Inferiority — Per ICH E14, an increase in the QTcF interval of 5 ms, as evidenced by the upper bound of a 95% one-sided confidence interval above 0.10, is the threshold for regulatory concern. Statistically, the test of prolongation is equivalent to a non-inferiority test versus placebo by crossover design, with an non-inferiority margin of 10 ms; Least-Squares Mean Double Delta Value = -0.99, 95% CI 1-sided [upper limit 0.635]
Statistical Analysis 2: Comparison: 2 g of Zoliflodacin vs Placebo; Null Hypothesis: Zoliflodacin administered at a 2 g dose causes a prolongation of the QTcF interval 1 h post-dose that exceeds the criteria in the ICH Guidance E14 (5 ms); Test type: Non-Inferiority — Per ICH E14, an increase in the QTcF interval of 5 ms, as evidenced by the upper bound of a 95% one-sided confidence interval above 0.10, is the threshold for regulatory concern; Least-Squares Mean Double Delta Value = 0.59, 95% CI 1-sided [upper limit 2.200]
Statistical Analysis 3: Comparison: 2 g of Zoliflodacin vs Placebo; Null Hypothesis: Zoliflodacin administered at a 2 g dose causes a prolongation of the QTcF interval 2 h post-dose that exceeds the criteria in the ICH Guidance E14 (5 ms); Test type: Non-Inferiority — [test comment as in outcome 1, analysis 2]; Least-Squares Mean Double Delta Value = 0.17, 95% CI 1-sided [upper limit 1.795]
Statistical Analysis 4: Comparison: 2 g of Zoliflodacin vs Placebo; Null Hypothesis: Zoliflodacin administered at a 2 g dose causes a prolongation of the QTcF interval 3 h post-dose that exceeds the criteria in the ICH Guidance E14 (5 ms); Test type: Non-Inferiority — [test comment as in outcome 1, analysis 2]; Least-Squares Mean Double Delta Value = 1.42, 95% CI 1-sided [upper limit 3.044]
Statistical Analysis 5: Comparison: 2 g of Zoliflodacin vs Placebo; Null Hypothesis: Zoliflodacin administered at a 2 g dose causes a prolongation of the QTcF interval 4 h post-dose that exceeds the criteria in the ICH Guidance E14 (5 ms); Test type: Non-Inferiority — [test comment as in outcome 1, analysis 2]; Least-Squares Mean Double Delta Value = 1.17, 95% CI 1-sided [upper limit 2.792]
Statistical Analysis 6: Comparison: 2 g of Zoliflodacin vs Placebo; Null Hypothesis: Zoliflodacin administered at a 2 g dose causes a prolongation of the QTcF interval 6 h post-dose that exceeds the criteria in the ICH Guidance E14 (5 ms); Test type: Non-Inferiority — [test comment as in outcome 1, analysis 2]; Least-Squares Mean Double Delta Value = 0.45, 95% CI 1-sided [upper limit 2.074]
Statistical Analysis 7: Comparison: 2 g of Zoliflodacin vs Placebo; Null Hypothesis: Zoliflodacin administered at a 2 g dose causes a prolongation of the QTcF interval 8 h post-dose that exceeds the criteria in the ICH Guidance E14 (5 ms); Test type: Non-Inferiority — [test comment as in outcome 1, analysis 2]; Least-Squares Mean Double Delta Value = -0.83, 95% CI 1-sided [upper limit 0.790]
Statistical Analysis 8: Comparison: 2 g of Zoliflodacin vs Placebo; Null Hypothesis: Zoliflodacin administered at a 2 g dose causes a prolongation of the QTcF interval 12 h post-dose that exceeds the criteria in the ICH Guidance E14 (5 ms); Test type: Non-Inferiority — [test comment as in outcome 1, analysis 2]; Least-Squares Mean Double Delta Value = 0.03, 95% CI 1-sided [upper limit 1.650]
Statistical Analysis 9: Comparison: 2 g of Zoliflodacin vs Placebo; Null Hypothesis: Zoliflodacin administered at a 2 g dose causes a prolongation of the QTcF interval 24 h post-dose that exceeds the criteria in the ICH Guidance E14 (5 ms); Test type: Non-Inferiority — [test comment as in outcome 1, analysis 2]; Least-Squares Mean Double Delta Value = -0.53, 95% CI 1-sided [upper limit 1.131]
Statistical Analysis 10: Comparison: 4 g of Zoliflodacin vs Placebo; Null Hypothesis: Zoliflodacin administered at a 4 g dose causes a prolongation of the QTcF interval 0.5 h post-dose that exceeds the criteria in the ICH Guidance E14 (5 ms); Test type: Non-Inferiority — [test comment as in outcome 1, analysis 2]; Least-Squares Mean Double Delta Value = 1.17, 95% CI 1-sided [upper limit 2.815]
Statistical Analysis 11: Comparison: 4 g of Zoliflodacin vs Placebo; Null Hypothesis: Zoliflodacin administered at a 4 g dose causes a prolongation of the QTcF interval 1 h post-dose that exceeds the criteria in the ICH Guidance E14 (5 ms); Test type: Non-Inferiority — [test comment as in outcome 1, analysis 2]; Least-Squares Mean Double Delta Value = 2.36, 95% CI 1-sided [upper limit 3.997]
Statistical Analysis 12: Comparison: 4 g of Zoliflodacin vs Placebo; Null Hypothesis: Zoliflodacin administered at a 4 g dose causes a prolongation of the QTcF interval 2 h post-dose that exceeds the criteria in the ICH Guidance E14 (5 ms); Test type: Non-Inferiority — [test comment as in outcome 1, analysis 2]; Least-Squares Mean Double Delta Value = 2.18, 95% CI 1-sided [upper limit 3.812]
Statistical Analysis 13: Comparison: 4 g of Zoliflodacin vs Placebo; Null Hypothesis: Zoliflodacin administered at a 4 g dose causes a prolongation of the QTcF interval 3 h post-dose that exceeds the criteria in the ICH Guidance E14 (5 ms); Test type: Non-Inferiority — [test comment as in outcome 1, analysis 2]; Least-Squares Mean Double Delta Value = 2.59, 95% CI 1-sided [upper limit 4.228]
Statistical Analysis 14: Comparison: 4 g of Zoliflodacin vs Placebo; Null Hypothesis: Zoliflodacin administered at a 4 g dose causes a prolongation of the QTcF interval 4 h post-dose that exceeds the criteria in the ICH Guidance E14 (5 ms); Test type: Non-Inferiority — [test comment as in outcome 1, analysis 2]; Least-Squares Mean Double Delta Value = 3.04, 95% CI 1-sided [upper limit 4.674]
Statistical Analysis 15: Comparison: 4 g of Zoliflodacin vs Placebo; Null Hypothesis: Zoliflodacin administered at a 4 g dose causes a prolongation of the QTcF interval 6 h post-dose that exceeds the criteria in the ICH Guidance E14 (5 ms); Test type: Non-Inferiority — [test comment as in outcome 1, analysis 2]; Least-Squares Mean Double Delta Value = 1.63, 95% CI 1-sided [upper limit 3.259]
Statistical Analysis 16: Comparison: 4 g of Zoliflodacin vs Placebo; Null Hypothesis: Zoliflodacin administered at a 4 g dose causes a prolongation of the QTcF interval 8 h post-dose that exceeds the criteria in the ICH Guidance E14 (5 ms); Test type: Non-Inferiority — [test comment as in outcome 1, analysis 2]; Least-Squares Mean Double Delta Value = -0.07, 95% CI 1-sided [upper limit 1.566]
Statistical Analysis 17: Comparison: 4 g of Zoliflodacin vs Placebo; Null Hypothesis: Zoliflodacin administered at a 4 g dose causes a prolongation of the QTcF interval 12 h post-dose that exceeds the criteria in the ICH Guidance E14 (5 ms); Test type: Non-Inferiority — [test comment as in outcome 1, analysis 2]; Least-Squares Mean Double Delta Value = 1.82, 95% CI 1-sided [upper limit 3.459]
Statistical Analysis 18: Comparison: 4 g of Zoliflodacin vs Placebo; Null Hypothesis: Zoliflodacin administered at a 4 g dose causes a prolongation of the QTcF interval 24 h post-dose that exceeds the criteria in the ICH Guidance E14 (5 ms); Test type: Non-Inferiority — [test comment as in outcome 1, analysis 2]; Least-Squares Mean Double Delta Value = 1.72, 95% CI 1-sided [upper limit 3.415]

2. Secondary Outcome: Time-matched, Placebo-corrected, Baseline-adjusted Heart Rate (HR) Following Administration of Zoliflodacin
Description: Mean and 90% two-sided confidence intervals (t-intervals) of change from baseline heart rate by time point and treatment. Note that the upper bound of the 90% two-sided confidence interval can also be interpreted as the upper bound of a 95% one-sided confidence interval.
Time Frame: Baseline, 0.5 h, 1 h, 2 h, 3 h, 4 h, 6 h, 8 h, 12 h, and 24 h post-dose
Population: The analysis population sample size is equal to the number of subjects in the Holter ECG Analysis Population who received both a dose of zoliflodacin and a dose of placebo.
Measure: Mean (95% Confidence Interval); unit: beats/minute
Arm/Group | 2 g of Zoliflodacin | 4 g of Zoliflodacin | Placebo
Number analyzed (Participants) | 68 | 66 | 69
beats/minute
  0.5 hour post dose: number analyzed (Participants) | 67 | 66 | 69
  0.5 hour post dose | 0.4 [-0.50 to 1.24] | 2.2 [1.36 to 2.94] | 0.1 [-0.50 to 0.77]
  1 hour post dose | 1.6 [0.60 to 2.55] | 2.3 [1.55 to 3.00] | -0.6 [-1.20 to 0.07]
  2 hour post dose | 1.0 [0.29 to 1.80] | 3.6 [2.24 to 5.01] | 0.1 [-0.62 to 0.82]
  3 hour post dose | 2.2 [1.35 to 3.00] | 4.5 [3.05 to 5.95] | 0.7 [-0.29 to 1.68]
  4 hour post dose | 1.6 [0.69 to 2.54] | 3.7 [2.32 to 5.04] | 0.00 [-0.85 to 0.94]
  6 hour post dose: number analyzed (Participants) | 67 | 66 | 69
  6 hour post dose | 9.4 [7.95 to 10.79] | 10.0 [8.40 to 11.54] | 7.8 [6.62 to 8.95]
  8 hour post dose | 8.7 [7.52 to 9.89] | 8.3 [6.86 to 9.84] | 5.8 [4.71 to 6.94]
  12 hour post dose: number analyzed (Participants) | 67 | 66 | 69
  12 hour post dose | 10.6 [9.13 to 12.00] | 10.4 [9.01 to 11.77] | 9.7 [8.37 to 10.96]
  24 hour post dose: number analyzed (Participants) | 68 | 65 | 66
  24 hour post dose | 2.5 [1.60 to 3.37] | 2.8 [1.66 to 3.85] | 3.4 [2.20 to 4.52]

3. Secondary Outcome: Time-matched, Placebo-corrected, Baseline-adjusted, the Time From the Onset of the P Wave to the Start of the QRS Complex (PR Interval) Following Administration of Zoliflodacin
Description: Mean and 90% two-sided confidence intervals (t-intervals) of change from baseline PR intervals by time point and treatment. Note that the upper bound of the 90% two-sided confidence interval can also be interpreted as the upper bound of a 95% one-sided confidence interval.
Time Frame: Baseline, 0.5 h, 1 h, 2 h, 3 h, 4 h, 6 h, 8 h, 12 h, and 24 h post-dose
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: milliseconds (msec)
Arm/Group | 2 g of Zoliflodacin | 4 g of Zoliflodacin | Placebo
Number analyzed (Participants) | 68 | 66 | 69
milliseconds (msec)
  0.5 hour post dose: number analyzed (Participants) | 67 | 65 | 69
  0.5 hour post dose | -0.7 [-1.90 to 0.53] | -1.1 [-2.01 to -0.24] | -0.3 [-1.35 to 0.74]
  1 hour post dose | -0.9 [-2.04 to 0.33] | -2.3 [-3.31 to -1.35] | 0.2 [-0.70 to 1.02]
  2 hour post dose: number analyzed (Participants) | 67 | 66 | 69
  2 hour post dose | -1.6 [-2.69 to -0.47] | -1.8 [-3.09 to -0.49] | -0.2 [-1.11 to 0.77]
  3 hour post dose: number analyzed (Participants) | 67 | 66 | 69
  3 hour post dose | -2.6 [-4.11 to -1.02] | -2.9 [-4.17 to -1.65] | -1.1 [-2.24 to -0.02]
  4 hour post dose: number analyzed (Participants) | 67 | 66 | 69
  4 hour post dose | -2.8 [-4.00 to -1.52] | -3.2 [-4.35 to -1.95] | -0.6 [-1.68 to 0.52]
  6 hour post dose: number analyzed (Participants) | 67 | 66 | 69
  6 hour post dose | -3.6 [-5.60 to -1.69] | -3.9 [-5.43 to -2.45] | -1.8 [-3.39 to -0.24]
  8 hour post dose: number analyzed (Participants) | 67 | 66 | 69
  8 hour post dose | -5.7 [-7.43 to -4.03] | -5.4 [-6.80 to -4.05] | -5.3 [-6.81 to -3.74]
  12 hour post dose: number analyzed (Participants) | 67 | 65 | 69
  12 hour post dose | -3.0 [-4.69 to -1.40] | -3.5 [-4.63 to -2.41] | -4.3 [-5.78 to -2.83]
  24 hour post dose: number analyzed (Participants) | 67 | 64 | 65
  24 hour post dose | -1.7 [-2.88 to -0.49] | -0.8 [-2.01 to 0.38] | -0.7 [-1.83 to 0.35]

4. Secondary Outcome: Time-matched, Placebo-corrected, Baseline-adjusted the Time Elapsed Between Two Successive R Waves of the QRS (RR Interval) Following Administration of Zoliflodacin
Description: Mean and 90% two-sided confidence intervals (t-intervals) of change from baseline RR intervals by time point and treatment. Note that the upper bound of the 90% two-sided confidence interval can also be interpreted as the upper bound of a 95% one-sided confidence interval.
Time Frame: Baseline, 0.5 h, 1 h, 2 h, 3 h, 4 h, 6 h, 8 h, 12 h, and 24 h post-dose
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: milliseconds (msec)
Arm/Group | 2 g of Zoliflodacin | 4 g of Zoliflodacin | Placebo
Number analyzed (Participants) | 68 | 66 | 69
milliseconds (msec)
  0.5 hour post dose: number analyzed (Participants) | 67 | 66 | 69
  0.5 hour post dose | -5.8 [-18.87 to 7.20] | -33.5 [-46.70 to -20.39] | -1.2 [-11.70 to 9.35]
  1 hour post dose | -22.6 [-36.30 to -8.81] | -35.0 [-46.45 to -23.58] | 9.7 [-0.72 to 20.08]
  2 hour post dose | -13.8 [-25.30 to -2.32] | -51.0 [-65.99 to -36.07] | 3.0 [-9.34 to 15.29]
  3 hour post dose | -32.0 [-43.54 to -20.52] | -63.1 [-80.01 to -46.21] | -10.1 [-24.26 to 4.00]
  4 hour post dose | -23.3 [-35.96 to -10.57] | -47.6 [-64.48 to -30.73] | -0.7 [-15.60 to 14.12]
  6 hour post dose: number analyzed (Participants) | 67 | 66 | 69
  6 hour post dose | -127.1 [-144.51 to -109.67] | -133.0 [-152.59 to -113.50] | -113.7 [-130.03 to -97.30]
  8 hour post dose | -120.2 [-135.53 to -104.88] | -111.0 [-127.57 to -94.37] | -87.5 [-102.32 to -72.75]
  12 hour post dose: number analyzed (Participants) | 67 | 66 | 69
  12 hour post dose | -141.2 [-159.18 to -123.21] | -139.8 [-155.48 to -124.06] | -140.5 [-159.15 to -121.78]
  24 hour post dose: number analyzed (Participants) | 68 | 65 | 66
  24 hour post dose | -37.4 [-49.72 to -25.05] | -41.2 [-57.11 to -25.25] | -50.2 [-65.39 to -35.06]

5. Secondary Outcome: Time-matched, Placebo-corrected, Baseline-adjusted QRS Duration Following Administration of Zoliflodacin
Description: Mean and 90% two-sided confidence intervals (t-intervals) of change from baseline QRS durations by time point and treatment. Note that the upper bound of the 90% two-sided confidence interval can also be interpreted as the upper bound of a 95% one-sided confidence interval.
Time Frame: Baseline, 0.5 h, 1 h, 2 h, 3 h, 4 h, 6 h, 8 h, 12 h, and 24 h post-dose
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: milliseconds (msec)
Arm/Group | 2 g of Zoliflodacin | 4 g of Zoliflodacin | Placebo
Number analyzed (Participants) | 68 | 66 | 69
milliseconds (msec)
  0.5 hour post dose: number analyzed (Participants) | 67 | 65 | 69
  0.5 hour post dose | -0.3 [-0.60 to 0.07] | -0.1 [-0.45 to 0.24] | -0.3 [-0.63 to -0.04]
  1 hour post dose | -0.5 [-0.87 to -0.16] | 0.1 [-0.23 to 0.38] | 0.0 [-0.28 to 0.34]
  2 hour post dose: number analyzed (Participants) | 67 | 66 | 69
  2 hour post dose | -0.6 [-0.91 to -0.25] | -0.5 [-0.90 to -0.20] | 0.0 [-0.47 to 0.47]
  3 hour post dose: number analyzed (Participants) | 67 | 66 | 69
  3 hour post dose | -0.4 [-0.70 to -0.08] | -0.4 [-0.72 to -0.07] | -0.1 [-0.35 to 0.23]
  4 hour post dose: number analyzed (Participants) | 67 | 66 | 69
  4 hour post dose | -0.5 [-0.82 to -0.19] | -0.2 [-0.57 to 0.12] | -0.1 [-0.50 to 0.21]
  6 hour post dose: number analyzed (Participants) | 67 | 66 | 69
  6 hour post dose | 0.1 [-0.34 to 0.49] | 0.1 [-0.25 to 0.49] | 0.8 [0.43 to 1.22]
  8 hour post dose: number analyzed (Participants) | 67 | 66 | 69
  8 hour post dose | -0.7 [-1.03 to -0.28] | -0.7 [-1.08 to -0.26] | -0.3 [-0.69 to 0.05]
  12 hour post dose: number analyzed (Participants) | 67 | 65 | 69
  12 hour post dose | -0.4 [-0.79 to 0.02] | -0.5 [-0.77 to -0.15] | -0.3 [-0.66 to 0.14]
  24 hour post dose: number analyzed (Participants) | 67 | 64 | 65
  24 hour post dose | -0.5 [-0.89 to -0.12] | -0.2 [-0.61 to 0.18] | -0.4 [-0.67 to -0.07]

6. Secondary Outcome: The One-sided 95% Confidence Interval (CI) of the Time-matched, Placebo-corrected, Baseline-adjusted Mean QTcF Interval (Delta Delta QTcF) After a Single Dose of Moxifloxacin
Description: as for outcome 1
Time Frame: Baseline, 1 h, 2 h, 3 h, and 4 h post-dose
Population: Any participants who received a dose of moxifloxacin and placebo and had post dose assessments is counted in the population.
Measure: Mean (95% Confidence Interval); unit: milliseconds (msec)
Groups:
- 400 mg of Moxifloxacin: 400 mg of moxifloxacin administered orally on Day 1 of dosing period.
- Placebo: Placebo administered orally on Day 1 of dosing period.
Arm/Group | 400 mg of Moxifloxacin | Placebo
Number analyzed (Participants) | 70 | 69
milliseconds (msec)
  1 hour post dose | 7.9 [6.81 to 8.99] | -2.3 [-3.34 to -1.29]
  2 hour post dose | 8.5 [7.32 to 9.59] | -2.2 [-3.30 to -1.19]
  3 hour post dose | 8.0 [6.67 to 9.36] | -2.6 [-3.78 to -1.32]
  4 hour post dose: number analyzed (Participants) | 69 | 69
  4 hour post dose | 7.2 [5.93 to 8.53] | -3.3 [-4.36 to -2.16]
Statistical Analysis 1: Comparison: 400 mg of Moxifloxacin vs Placebo; Null Hypothesis: The trial does not have the sensitivity to detect an effect on QTcF of regulatory concern, as produced by 400 mg moxifloxacin 1 h after dose; Test type: Non-Inferiority — According to ICH E14, "the positive control should have an effect on the mean QT/QTc interval of about 5 ms." Comparison of the lower bound of the confidence interval to 5 ms for a 400 mg dose of moxifloxacin is standard practice for demonstrating assay sensitivity in thorough QT studies; Least-Squares Mean Double Delta Value = 10.19, 98.75% CI 1-sided [lower limit 8.257]
Statistical Analysis 2: Comparison: 400 mg of Moxifloxacin vs Placebo; Null Hypothesis: The trial does not have the sensitivity to detect an effect on QTcF of regulatory concern, as produced by 400 mg moxifloxacin 2 h after dose; Test type: Non-Inferiority — [test comment as in outcome 6, analysis 1]; Least-Squares Mean Double Delta Value = 10.79, 98.75% CI 1-sided [lower limit 8.860]
Statistical Analysis 3: Comparison: 400 mg of Moxifloxacin vs Placebo; Null Hypothesis: The trial does not have the sensitivity to detect an effect on QTcF of regulatory concern, as produced by 400 mg moxifloxacin 3 h after dose; Test type: Non-Inferiority — [test comment as in outcome 6, analysis 1]; Least-Squares Mean Double Delta Value = 10.62, 98.75% CI 1-sided [lower limit 8.683]
Statistical Analysis 4: Comparison: 400 mg of Moxifloxacin vs Placebo; Null Hypothesis: The trial does not have the sensitivity to detect an effect on QTcF of regulatory concern, as produced by 400 mg moxifloxacin 4 h after dose; Test type: Non-Inferiority — [test comment as in outcome 6, analysis 1]; Least-Squares Mean Double Delta Value = 10.63, 98.75% CI 1-sided [lower limit 8.698]

7. Secondary Outcome: Incidence of Abnormal T-wave Morphology Following Administration of Zoliflodacin
Description: Categorical T-wave morphology analysis was collected in three ECG replicates at each timepoint (Baseline, 0.5 h, 1 h, 2 h, 3 h, 4 h, 6 h, 8 h, 12 h, and 24 h post-dose). Abnormalities present in any one or more of the baseline timepoint replicate ECGs recorded for a particular period was considered to be present at baseline for post-dose ECGs from that specific period. If a subject had an ECG morphological abnormality in more than one replicate ECG of a study timepoint, the subject was counted only once for that timepoint. Flat is defined as T amplitude <1 mm (either positive or negative) including flat isoelectric line and Biphasic is defined as T-wave that contains a second component with an opposite phase that was at least 0.1 millivolts (mV) deep (both positive and negative/positive and polyphasic T-waves included).
Time Frame: Baseline, 0.5 h, 1 h, 2 h, 3 h, 4 h, 6 h, 8 h, 12 h, and 24 h post-dose
Population: Any participants who received study product and had post dose assessments.
Measure: Count of Participants; unit: Participants
Groups:
- Placebo: Placebo for zoliflodacin administered orally on Day 1 of each dosing period
  Placebo: Composed of 4g of the same excipients found in zoliflodacin. Powder was reconstituted in 60 mL of water and dosed orally. After the cup containing 60 mL of placebo was taken, approximately 60 mL of water was consumed by the subject to chase the initial dose.
- 2 g of Zoliflodacin: 2 g of zoliflodacin administered orally on Day 1 of each dosing period
  AZD0914: Spiropyrimidinetrione antibacterial drug, powder (zoliflodacin) was reconstituted in 60 mL of water and dosed orally following an overnight fast, after which approximately 60 mL of water was added to the cup and consumed by the subject.
- 4 g of Zoliflodacin: 4 g of zoliflodacin administered orally on Day 1 of each dosing period
  AZD0914: Spiropyrimidinetrione antibacterial drug, powder (zoliflodacin) was reconstituted in 60 mL of water and dosed orally following an overnight fast, after which approximately 60 mL of water was added to the cup and consumed by the subject.
- 400 mg of Moxifloxacin: 400 mg of moxifloxacin administered orally on Day 1 of each dosing period
  Moxifloxacin: Broad-spectrum 8-methoxy fluoroquinolone. A single, commercially-available, film-coated, 400-mg tablet of moxifloxacin hydrochloride was administered orally with 120 mL of water.
Arm/Group | Placebo | 2 g of Zoliflodacin | 4 g of Zoliflodacin | 400 mg of Moxifloxacin
Number analyzed (Participants) | 69 | 68 | 66 | 70
Participants
  0.5 h post dose: T wave: Abnormal, Biphasic | 0 | 0 | 0 | 0
  0.5 h post dose: T wave: Abnormal, Flat | 0 | 0 | 0 | 0
  0.5 h post: T wave:Abnormal, Inverted, Asymmetric | 0 | 0 | 0 | 0
  1 h post dose: T wave: Abnormal, Biphasic | 0 | 0 | 0 | 0
  1 h post dose: T wave: Abnormal, Flat | 0 | 0 | 0 | 0
  1 h post: T wave: Abnormal, Inverted, Asymmetric | 0 | 0 | 0 | 0
  2 h post dose: T wave: Abnormal, Biphasic | 0 | 0 | 0 | 0
  2 h post dose: T wave: Abnormal, Flat | 0 | 0 | 2 | 1
  2 h post: T wave: Abnormal, Inverted, Asymmetric | 0 | 0 | 0 | 0
  3 h post dose: T wave: Abnormal, Biphasic | 0 | 0 | 0 | 0
  3 h post dose: T wave: Abnormal, Flat | 0 | 0 | 2 | 0
  3 h post:T wave: Abnormal, Inverted, Asymmetric | 0 | 0 | 1 | 0
  4 h post dose: T wave: Abnormal, Biphasic: number analyzed (Participants) | 69 | 68 | 66 | 69
  4 h post dose: T wave: Abnormal, Biphasic | 0 | 0 | 0 | 0
  4 h post dose: T wave: Abnormal, Flat: number analyzed (Participants) | 69 | 68 | 66 | 69
  4 h post dose: T wave: Abnormal, Flat | 0 | 0 | 2 | 0
  4 h post:T wave: Abnormal, Inverted, Asymmetric: number analyzed (Participants) | 69 | 68 | 66 | 69
  4 h post:T wave: Abnormal, Inverted, Asymmetric | 0 | 0 | 1 | 0
  6 h post dose: T wave: Abnormal, Biphasic: number analyzed (Participants) | 69 | 68 | 66 | 69
  6 h post dose: T wave: Abnormal, Biphasic | 0 | 0 | 1 | 0
  6 h post dose: T wave: Abnormal, Flat: number analyzed (Participants) | 69 | 68 | 66 | 69
  6 h post dose: T wave: Abnormal, Flat | 6 | 4 | 4 | 5
  6 h post:T wave: Abnormal, Inverted, Asymmetric: number analyzed (Participants) | 69 | 68 | 66 | 69
  6 h post:T wave: Abnormal, Inverted, Asymmetric | 2 | 0 | 1 | 1
  8 h post dose: T wave: Abnormal, Biphasic: number analyzed (Participants) | 69 | 68 | 66 | 69
  8 h post dose: T wave: Abnormal, Biphasic | 0 | 0 | 1 | 0
  8 h post dose: T wave: Abnormal, Flat: number analyzed (Participants) | 69 | 68 | 66 | 69
  8 h post dose: T wave: Abnormal, Flat | 3 | 1 | 2 | 1
  8 h post:T wave: Abnormal, Inverted, Asymmetric: number analyzed (Participants) | 69 | 68 | 66 | 69
  8 h post:T wave: Abnormal, Inverted, Asymmetric | 0 | 0 | 1 | 0
  12 h post dose: T wave: Abnormal, Biphasic: number analyzed (Participants) | 69 | 68 | 66 | 69
  12 h post dose: T wave: Abnormal, Biphasic | 0 | 0 | 1 | 0
  12 h post dose: T wave: Abnormal, Flat: number analyzed (Participants) | 69 | 68 | 66 | 69
  12 h post dose: T wave: Abnormal, Flat | 1 | 4 | 2 | 1
  12 h post:T wave: Abnormal, Inverted, Asymmetric: number analyzed (Participants) | 69 | 68 | 66 | 69
  12 h post:T wave: Abnormal, Inverted, Asymmetric | 0 | 1 | 1 | 0
  24 h post dose: T wave: Abnormal, Biphasic: number analyzed (Participants) | 66 | 68 | 65 | 69
  24 h post dose: T wave: Abnormal, Biphasic | 0 | 0 | 1 | 0
  24 h post dose: T wave: Abnormal, Flat: number analyzed (Participants) | 66 | 68 | 65 | 69
  24 h post dose: T wave: Abnormal, Flat | 0 | 0 | 0 | 1
  24 h post:T wave: Abnormal, Inverted, Asymmetric: number analyzed (Participants) | 66 | 68 | 65 | 69
  24 h post:T wave: Abnormal, Inverted, Asymmetric | 0 | 0 | 0 | 0

8. Secondary Outcome: Maximum Observed Concentration (Cmax) of Zoliflodacin
Description: Cmax is defined as the maximum observed drug concentration observed in plasma over all PK sample concentrations computed from concentrations that were measured using a validated HPLC-MS/MS method. Pharmacokinetic (PK) parameters were computed using plasma concentrations from samples collected pre-dose and intervals post-dose.
Time Frame: Baseline, 0.5 h, 1 h, 2 h, 3 h, 4 h, 6 h, 8 h, 12 h, and 24 h post-dose
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | 2 g of Zoliflodacin | 4 g of Zoliflodacin
Number analyzed (Participants) | 69 | 67
ng/mL | 12120 (2985) | 20350 (8682)

9. Secondary Outcome: Time of Maximum Observed Concentration (Tmax) of Zoliflodacin
Description: Tmax is defined as the time at which the maximum concentration (Cmax) occurs in plasma computed from concentrations that were measured using a validated HPLC-MS/MS method. PK parameters were computed using plasma concentrations from samples collected pre-dose and intervals post-dose.
Time Frame: Baseline, 0.5 h, 1 h, 2 h, 3 h, 4 h, 6 h, 8 h, 12 h, and 24 h post-dose
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | 2 g of Zoliflodacin | 4 g of Zoliflodacin
Number analyzed (Participants) | 69 | 67
hour | 2.90 (1.08) | 3.03 (2.05)

10. Secondary Outcome: Area Under the Concentration Time-curve From Time Zero to Infinity (AUC(0 - Infinity)) for Zoliflodacin
Description: AUC(0 - infinity) was defined as the total area under the concentration-time curve from dosing (time 0) taken to the limit as the end time becomes arbitrarily large. AUC(0 - infinity) was calculated by adding AUC(0-last) to an extrapolated value equal to the last measured concentration greater than the lower limit of quantification of the bioanalytical assay divided by the terminal phase elimination rate constant (Ke) computed from concentrations that were measured using a validated HPLC-MS/MS method. PK parameters were computed using plasma concentrations from samples collected pre-dose and intervals post-dose.
Time Frame: Baseline, 0.5 h, 1 h, 2 h, 3 h, 4 h, 6 h, 8 h, 12 h, and 24 h post-dose
Measure: Mean (Standard Deviation); unit: h x ng/mL
Arm/Group | 2 g of Zoliflodacin | 4 g of Zoliflodacin
Number analyzed (Participants) | 69 | 67
h x ng/mL | 108300 (32980) | 181400 (52890)

11. Secondary Outcome: Area Under the Concentration Time-curve From Time Zero to the Last Concentration Above the Lower Limit of Quantitation (AUC(0-last)) for Zoliflodacin
Description: AUC(0-last) was defined as the area under the concentration-time curve from dosing (time 0) to the time of the last measured concentration computed from concentrations that were measured using a validated HPLC-MS/MS method. PK parameters were computed using plasma concentrations from samples collected pre-dose and intervals post-dose.
Time Frame: Baseline, 0.5 h, 1 h, 2 h, 3 h, 4 h, 6 h, 8 h, 12 h, and 24 h post-dose
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | 2 g of Zoliflodacin | 4 g of Zoliflodacin
Number analyzed (Participants) | 69 | 67
h*ng/mL | 102700 (28580) | 177300 (52370)

12. Secondary Outcome: Apparent Volume of Distribution (Vz/F) of Zoliflodacin
Description: Apparent volume of distribution during terminal phase (Vz/F) after non-intravenous administration was calculated as (CL/F)/ Ke computed from concentrations that were measured using a validated HPLC-MS/MS method. PK parameters were computed using plasma concentrations from samples collected pre-dose and intervals post-dose.
Time Frame: Baseline, 0.5 h, 1 h, 2 h, 3 h, 4 h, 6 h, 8 h, 12 h, and 24 h post-dose
Measure: Mean (Standard Deviation); unit: Liter
Arm/Group | 2 g of Zoliflodacin | 4 g of Zoliflodacin
Number analyzed (Participants) | 50 | 42
Liter | 160.55 (50.46) | 204.29 (55.13)

13. Secondary Outcome: Apparent Oral Clearance (CL/F) of Zoliflodacin
Description: Apparent oral clearance (CL/F) computed as Dose/Area under the curve (AUC) from time zero to infinity (0-infinity) computed from concentrations that were measured using a validated high-performance liquid chromatography-tandem mass spectrometry (HPLC-MS/MS) method. PK parameters were computed using plasma concentrations from samples collected pre-dose and intervals post-dose.
Time Frame: Baseline, 0.5 h, 1 h, 2 h, 3 h, 4 h, 6 h, 8 h, 12 h, and 24 h post-dose
Measure: Mean (Standard Deviation); unit: Liter/hour
Arm/Group | 2 g of Zoliflodacin | 4 g of Zoliflodacin
Number analyzed (Participants) | 50 | 42
Liter/hour | 20.08 (5.74) | 23.77 (6.34)

14. Secondary Outcome: Elimination Rate Constant (Ke) of Zoliflodacin
Description: The terminal phase elimination rate constant (Ke) was defined as the first-order rate constant describing the rate of decrease of drug concentration in the terminal phase (defined as the terminal region of the PK curve where drug concentration follows first-order elimination kinetics) computed from concentrations that were measured using a validated HPLC-MS/MS method. PK parameters were computed using plasma concentrations from samples collected pre-dose and intervals post-dose.
Time Frame: Baseline, 0.5 h, 1 h, 2 h, 3 h, 4 h, 6 h, 8 h, 12 h, and 24 h post-dose
Measure: Mean (Standard Deviation); unit: 1/hour
Arm/Group | 2 g of Zoliflodacin | 4 g of Zoliflodacin
Number analyzed (Participants) | 50 | 42
1/hour | 0.1267 (0.01590) | 0.1174 (0.01467)

15. Secondary Outcome: Terminal Elimination Half-life (t1/2) of Zoliflodacin
Description: The apparent terminal elimination half-life (t1/2) was defined as the time required for the drug concentration to decrease by a factor of one-half in the terminal phase computed from concentrations that were measured using a validated HPLC-MS/MS method. PK parameters were computed using plasma concentrations from samples collected pre-dose and intervals post-dose.
Time Frame: Baseline, 0.5 h, 1 h, 2 h, 3 h, 4 h, 6 h, 8 h, 12 h, and 24 h post-dose
Measure: Mean (Standard Deviation); unit: Hour
Arm/Group | 2 g of Zoliflodacin | 4 g of Zoliflodacin
Number analyzed (Participants) | 50 | 42
Hour | 5.55 (0.67) | 5.99 (0.71)

16. Secondary Outcome: Relationship Between Plasma Concentrations of Zoliflodacin and Time-matched, Placebo-corrected, Baseline-adjusted Mean QTcF Interval (Delta Delta QTcF) Following Administration of Zoliflodacin
Description: One-sided 95% confidence intervals of population mean QTcF time-matched, placebo-corrected, baseline-adjusted mean QTcF interval at plasma concentration corresponding to the observed geometric mean Cmax for 2 g and 4 g doses of zoliflodacin were computed using a linear mixed effect model with PK and concentration data collected at baseline and intervals post-dose.
Time Frame: Baseline, 0.5 h, 1 h, 2 h, 3 h, 4 h, 6 h, 8 h, 12 h, and 24 h post-dose
Population: Any participants who received study product and had post dose assessments.
Measure: Mean (95% Confidence Interval); unit: milliseconds (msec)
Arm/Group | 2 g of Zoliflodacin | 4 g of Zoliflodacin
Number analyzed (Participants) | 67 | 65
milliseconds (msec) | 1.5 [NA to 2.54] — The NA values shown in the lower bounds are a stand-in for negative infinity (-8). | 3.0 [NA to 4.41] — The NA values shown in the lower bounds are a stand-in for negative infinity (-8).

17. Secondary Outcome: Number of Participants With Treatment-emergent Serious Adverse Events Following Administration of Zoliflodacin and Moxifloxacin
Description: Serious adverse events included any untoward medical occurrence that resulted in death; was life threatening; was a persistent/significant disability/incapacity; required inpatient hospitalization or prolongation or a congenital anomaly/birth defect.
Time Frame: From study product administration (Day 1) through prior to the next dose (Day 8 or Final visit).
Population: Any participants who received study product.
Measure: Count of Participants; unit: Participants
Arm/Group | 2 g of Zoliflodacin | 4 g of Zoliflodacin | Placebo | 400 mg of Moxifloxacin
Number analyzed (Participants) | 69 | 67 | 70 | 71
Participants | 0 | 0 | 0 | 0

18. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events Following Administration of Study Product
Description: Adverse events are defined as any untoward medical occurrence regardless of its causal relationship to the study treatment.
Time Frame: From study product administration (Day 1) through prior to the next dose (Day 8 or Final visit).
Population: Any participants who received study product.
Measure: Count of Participants; unit: Participants
Arm/Group | 2 g of Zoliflodacin | 4 g of Zoliflodacin | Placebo | 400 mg of Moxifloxacin
Number analyzed (Participants) | 69 | 67 | 70 | 71
Participants | 38 | 46 | 35 | 41

19. Secondary Outcome: Changes From Baseline for Blood Pressure - Systolic
Description: Change from baseline in systolic blood pressure was calculated by subtracting the baseline (pre-dose) measurement from the post-dose measurement. Post-dose measurements were taken 1 h, 2 h, 4 h and 24 h after dosing. Follow up is defined as the check in visit for the next dosing period or the final visit.
Time Frame: From study product administration (Day 1) through prior to the next dose (Day 8 or Final visit).
Population: Any participants who received study product and had post dose assessments.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | 2 g of Zoliflodacin | 4 g of Zoliflodacin | Placebo | 400 mg of Moxifloxacin
Number analyzed (Participants) | 69 | 67 | 70 | 71
mmHg
  1 hour post dose | 0.8 (7.3) | 1.3 (7.9) | 0.8 (7.6) | 0.4 (7.8)
  2 hour post dose | 0.4 (8.0) | -0.3 (7.6) | 1.0 (8.6) | -0.5 (6.8)
  4 hour post dose: number analyzed (Participants) | 69 | 67 | 70 | 70
  4 hour post dose | 0.1 (7.1) | -0.9 (7.5) | 1.0 (7.6) | -1.7 (7.7)
  24 hour post dose: number analyzed (Participants) | 69 | 67 | 70 | 70
  24 hour post dose | 0.0 (8.2) | -0.4 (7.8) | 1.1 (7.3) | 0.5 (6.9)
  Follow up: number analyzed (Participants) | 68 | 67 | 67 | 69
  Follow up | 3.5 (8.2) | 2.3 (6.9) | 3.7 (9.2) | 5.0 (8.4)

20. Secondary Outcome: Changes From Baseline for Blood Pressure - Diastolic
Description: Change from baseline in diastolic blood pressure was calculated by subtracting the baseline (pre-dose) measurement from the post-dose measurement. Post-dose measurements were taken 1 h, 2 h, 4 h and 24 h after dosing. Follow up is defined as the check in visit for the next dosing period or the final visit.
Time Frame: From study product administration (Day 1) through prior to the next dose (Day 8 or Final visit).
Population: Any participants who received study product and had post dose assessments.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | 2 g of Zoliflodacin | 4 g of Zoliflodacin | Placebo | 400 mg of Moxifloxacin
Number analyzed (Participants) | 69 | 67 | 70 | 71
mmHg
  1 hour post dose | 0.3 (5.3) | 0.3 (4.8) | 0.8 (6.1) | 1.5 (5.3)
  2 hour post dose | -0.4 (6.0) | -0.9 (5.1) | 0.6 (6.7) | 1.2 (5.5)
  4 hour post dose: number analyzed (Participants) | 69 | 67 | 70 | 70
  4 hour post dose | -0.4 (4.9) | -2.3 (5.3) | 1.1 (5.7) | -0.1 (5.5)
  24 hour post dose: number analyzed (Participants) | 69 | 67 | 70 | 70
  24 hour post dose | 0.2 (5.3) | -0.5 (5.7) | 1.4 (5.4) | 1.1 (5.5)
  Follow up: number analyzed (Participants) | 68 | 67 | 67 | 69
  Follow up | 2.2 (5.3) | 0.5 (5.5) | 2.7 (6.7) | 3.8 (7.2)

21. Secondary Outcome: Changes From Baseline for Pulse Rate
Description: Change from baseline in pulse rate was calculated by subtracting the baseline (pre-dose) measurement from the post-dose measurement. Post-dose measurements were taken 1 h, 2 h, 4 h and 24 h after dosing. Follow up is defined as the check in visit for the next dosing period or the final visit.
Time Frame: From study product administration (Day 1) through prior to the next dose (Day 8 or Final visit).
Population: Any participants who received study product and had post dose assessments.
Measure: Mean (Standard Deviation); unit: beats/minute
Arm/Group | 2 g of Zoliflodacin | 4 g of Zoliflodacin | Placebo | 400 mg of Moxifloxacin
Number analyzed (Participants) | 69 | 67 | 70 | 71
beats/minute
  1 hour post dose | 5.2 (8.3) | 5.7 (7.8) | 2.8 (8.1) | 6.9 (6.8)
  2 hour post dose | 3.9 (7.8) | 6.5 (8.0) | 3.8 (7.5) | 5.5 (5.8)
  4 hour post dose: number analyzed (Participants) | 69 | 67 | 70 | 70
  4 hour post dose | 5.4 (8.5) | 5.8 (8.3) | 3.0 (9.6) | 5.2 (8.2)
  24 hour post dose: number analyzed (Participants) | 69 | 67 | 70 | 70
  24 hour post dose | 4.9 (7.7) | 5.2 (7.3) | 5.4 (8.4) | 6.3 (8.1)
  Follow up: number analyzed (Participants) | 68 | 67 | 67 | 69
  Follow up | 2.0 (8.7) | 2.8 (7.7) | 2.0 (10.3) | 4.2 (7.2)

22. Secondary Outcome: Changes From Baseline for Respiratory Rate
Description: Change from baseline in respiratory rate was calculated by subtracting the baseline (pre-dose) measurement from the post-dose measurement. Post-dose measurements were taken 1 h, 2 h, 4 h and 24 h after dosing. Follow up is defined as the check in visit for the next dosing period or the final visit.
Time Frame: From study product administration (Day 1) through prior to the next dose (Day 8 or Final visit).
Population: Any participants who received study product and had post dose assessments.
Measure: Mean (Standard Deviation); unit: breaths/minute
Arm/Group | 2 g of Zoliflodacin | 4 g of Zoliflodacin | Placebo | 400 mg of Moxifloxacin
Number analyzed (Participants) | 69 | 67 | 70 | 71
breaths/minute
  1 hour post dose: number analyzed (Participants) | 69 | 67 | 69 | 70
  1 hour post dose | 0.8 (3.1) | 1.1 (2.9) | 1.0 (2.8) | 0.4 (3.0)
  2 hour post dose | 0.4 (3.2) | 0.7 (2.9) | -0.3 (3.0) | 0.0 (3.0)
  4 hour post dose: number analyzed (Participants) | 69 | 67 | 70 | 70
  4 hour post dose | 0.8 (3.6) | 1.3 (3.3) | -0.2 (2.7) | 0.1 (3.1)
  24 hour post dose: number analyzed (Participants) | 69 | 67 | 70 | 70
  24 hour post dose | 0.9 (3.1) | 1.0 (2.9) | 0.6 (2.7) | 0.5 (3.0)
  Follow up: number analyzed (Participants) | 68 | 67 | 67 | 69
  Follow up | 0.6 (3.1) | 1.3 (3.3) | 0.2 (3.0) | 0.6 (3.6)

23. Secondary Outcome: Changes From Baseline for Temperature
Description: Change from baseline for temperature was calculated by subtracting the baseline (pre-dose) measurement from the post-dose measurement. Post-dose measurements were taken 1 h, 2 h, 4 h and 24 h after dosing. Follow up is defined as the check in visit for the next dosing period or the final visit.
Time Frame: From study product administration (Day 1) through prior to the next dose (Day 8 or Final visit).
Population: Any participants who received study product and had post dose assessments.
Measure: Mean (Standard Deviation); unit: Celsius
Arm/Group | 2 g of Zoliflodacin | 4 g of Zoliflodacin | Placebo | 400 mg of Moxifloxacin
Number analyzed (Participants) | 69 | 67 | 70 | 71
Celsius
  1 hour post dose | 0.08 (0.26) | 0.03 (0.25) | 0.03 (0.27) | 0.05 (0.31)
  2 hour post dose: number analyzed (Participants) | 69 | 66 | 69 | 71
  2 hour post dose | 0.10 (0.21) | 0.06 (0.22) | 0.09 (0.24) | 0.11 (0.23)
  4 hour post dose: number analyzed (Participants) | 69 | 67 | 70 | 70
  4 hour post dose | 0.08 (0.23) | 0.05 (0.27) | 0.09 (0.24) | 0.13 (0.26)
  24 hour post dose: number analyzed (Participants) | 69 | 67 | 70 | 70
  24 hour post dose | 0.09 (0.27) | 0.06 (0.27) | 0.04 (0.27) | 0.10 (0.26)
  Follow up: number analyzed (Participants) | 68 | 67 | 66 | 69
  Follow up | 0.05 (0.28) | -0.02 (0.31) | 0.00 (0.28) | 0.05 (0.29)

24. Secondary Outcome: Changes From Baseline for White Blood Cells With Differentials
Description: Change from baseline calculated by subtracting the Day -1 (baseline) hematology measurement from the 24 h post dose, and a follow up hematology measurement. Follow up is defined as either the check-in visit for the next period or the final visit. Hematology parameters included white blood cell count, and differential (absolute counts of neutrophils, lymphocytes, monocytes, eosinophils, and basophils).
Time Frame: Prior to dosing, 24 hour post dose through prior to the next dose (Day 8 or Final visit).
Population: Any participants who received study product and had post dose laboratory assessments.
Measure: Mean (Standard Deviation); unit: cells/microliter
Arm/Group | 2 g of Zoliflodacin | 4 g of Zoliflodacin | Placebo | 400 mg of Moxifloxacin
Number analyzed (Participants) | 69 | 67 | 70 | 70
cells/microliter
  Leukocytes: 24 hour post dose | -246.4 (1031.5) | -129.9 (1249.6) | -64.3 (1130.2) | -282.9 (1075.4)
  Leukocytes: Follow up: number analyzed (Participants) | 68 | 67 | 67 | 69
  Leukocytes: Follow up | -273.5 (1253.1) | 140.3 (1486.1) | 35.8 (1153.9) | -84.1 (1477.6)
  Neutrophils: 24 hour post dose | -248.0 (667.7) | -39.6 (955.3) | -54.3 (1036.5) | -351.3 (1008.5)
  Neutrophils: Follow up: number analyzed (Participants) | 68 | 67 | 67 | 69
  Neutrophils: Follow up | -272.2 (945.4) | 220.4 (1136.7) | -36.1 (986.4) | -59.2 (1216.6)
  Lymphocytes: 24 hour post dose | 3.4 (583.2) | -77.9 (499.6) | -1.9 (549.7) | 79.4 (556.9)
  Lymphocytes: Follow up: number analyzed (Participants) | 68 | 67 | 67 | 69
  Lymphocytes: Follow up | -19.6 (497.9) | -74.1 (530.5) | 96.9 (482.9) | -33.7 (625.8)
  Monocytes: 24 hour post dose | -7.8 (118.2) | -13.9 (125.3) | -10.6 (123.7) | -16.1 (114.8)
  Monocytes: Follow up: number analyzed (Participants) | 68 | 67 | 67 | 69
  Monocytes: Follow up | 4.6 (118.8) | -7.6 (158.7) | -25.4 (141.0) | 5.2 (138.9)
  Eosinophils: 24 hour post dose | 9.4 (65.1) | 4.0 (71.0) | 6.0 (72.8) | 8.2 (64.7)
  Eosinophils: Follow up: number analyzed (Participants) | 68 | 67 | 67 | 69
  Eosinophils: Follow up | 12.9 (80.9) | 2.2 (83.9) | 0.7 (69.7) | 2.3 (61.2)
  Basophils: 24 hour post dose | -3.4 (13.8) | -2.5 (13.3) | -3.3 (13.5) | -3.1 (14.4)
  Basophils: Follow up: number analyzed (Participants) | 68 | 67 | 67 | 69
  Basophils: Follow up | 0.6 (15.7) | -0.5 (14.9) | -0.2 (10.7) | 1.4 (14.7)

25. Secondary Outcome: Changes From Baseline for Hemoglobin
Description: Change from baseline for hemoglobin is calculated by subtracting the Day -1 (baseline) hematology measurement from the 24 h post dose, and a follow up hematology measurement. Follow up is defined as either the check-in visit for the next period or the final visit.
Time Frame: Prior to dosing, 24 hour post dose through prior to the next dose (Day 8 or Final visit).
Population: Any participants who received study product and had post dose laboratory assessments.
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | 2 g of Zoliflodacin | 4 g of Zoliflodacin | Placebo | 400 mg of Moxifloxacin
Number analyzed (Participants) | 69 | 67 | 70 | 70
g/dL
  Hemoglobin: 24 hour post dose | 0.15 (0.71) | 0.01 (0.65) | 0.04 (0.67) | -0.06 (0.68)
  Hemoglobin: Follow up: number analyzed (Participants) | 68 | 67 | 67 | 69
  Hemoglobin: Follow up | -0.01 (0.72) | -0.23 (0.68) | -0.06 (0.64) | -0.13 (0.70)

26. Secondary Outcome: Changes From Baseline for Hematocrit
Description: Change from baseline for hematocrit is calculated by subtracting the Day -1 (baseline) hematology measurement from the 24 h post dose, and a follow up hematology measurement. Follow up is defined as either the check-in visit for the next period or the final visit.
Time Frame: Prior to dosing, 24 hour post dose through prior to the next dose (Day 8 or Final visit).
Population: Any participants who received study product and had post dose laboratory assessments.
Measure: Mean (Standard Deviation); unit: volume percentage of RBC in blood
Arm/Group | 2 g of Zoliflodacin | 4 g of Zoliflodacin | Placebo | 400 mg of Moxifloxacin
Number analyzed (Participants) | 69 | 67 | 70 | 70
volume percentage of RBC in blood
  Hematocrit: 24 hour post dose | 0.39 (2.04) | -0.10 (2.02) | 0.08 (2.08) | -0.26 (2.13)
  Hematocrit: Follow up: number analyzed (Participants) | 68 | 67 | 67 | 69
  Hematocrit: Follow up | -0.03 (2.26) | -0.69 (2.15) | -0.10 (1.90) | -0.33 (2.19)

27. Secondary Outcome: Changes From Baseline for Erythrocytes
Description: Change from baseline for erythrocytes is calculated by subtracting the Day -1 (baseline) hematology measurement from the 24 h post dose, and a follow up hematology measurement. Follow up is defined as either the check-in visit for the next period or the final visit.
Time Frame: Prior to dosing, 24 hour post dose through prior to the next dose (Day 8 or Final visit).
Population: Any participants who received study product and had post dose laboratory assessments.
Measure: Mean (Standard Deviation); unit: 10^6 cells/microliter
Arm/Group | 2 g of Zoliflodacin | 4 g of Zoliflodacin | Placebo | 400 mg of Moxifloxacin
Number analyzed (Participants) | 69 | 67 | 70 | 70
10^6 cells/microliter
  Erythrocytes: 24 hour post dose | 0.050 (0.243) | -0.008 (0.228) | -0.002 (0.233) | -0.031 (0.253)
  Erythrocytes: Follow up: number analyzed (Participants) | 68 | 67 | 67 | 69
  Erythrocytes: Follow up | -0.005 (0.280) | -0.088 (0.249) | -0.029 (0.212) | -0.053 (0.248)

28. Secondary Outcome: Changes From Baseline for Platelets
Description: Change from baseline for platelets is calculated by subtracting the Day -1 (baseline) hematology measurement from the 24 h post dose, and a follow up hematology measurement. Follow up is defined as either the check-in visit for the next period or the final visit.
Time Frame: Prior to dosing, 24 hour post dose through prior to the next dose (Day 8 or Final visit).
Population: Any participants who received study product for that dosing period and had post dose laboratory assessments.
Measure: Mean (Standard Deviation); unit: 10^3 platelets/microliter
Arm/Group | 2 g of Zoliflodacin | 4 g of Zoliflodacin | Placebo | 400 mg of Moxifloxacin
Number analyzed (Participants) | 69 | 67 | 70 | 70
10^3 platelets/microliter
  Platelets: 24 hour post dose | -8.2 (25.8) | -10.3 (26.9) | -10.5 (24.4) | -15.4 (23.3)
  Platelets: Follow up: number analyzed (Participants) | 68 | 67 | 67 | 69
  Platelets: Follow up | 1.7 (27.8) | 2.9 (30.4) | 6.2 (30.3) | -3.8 (29.3)

29. Secondary Outcome: Changes From Baseline for Sodium, Potassium, Chloride and Bicarbonate
Description: Change from baseline calculated by subtracting the Day -1 (baseline) chemistry measurement from the 24 h post dose, and a follow up chemistry measurement. Follow up is defined as either the check-in visit for the next period or the final visit. Chemistry parameters included sodium, potassium. chloride and bicarbonate.
Time Frame: Prior to dosing, 24 hour post dose through prior to the next dose (Day 8 or Final visit).
Population: Any participants who received study product for that dosing period and had post dose laboratory assessments.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | 2 g of Zoliflodacin | 4 g of Zoliflodacin | Placebo | 400 mg of Moxifloxacin
Number analyzed (Participants) | 69 | 67 | 70 | 70
mmol/L
  Sodium: 24 hour post dose | 0.2 (1.9) | -0.1 (1.9) | 0.6 (1.9) | 0.7 (1.9)
  Sodium: Follow up: number analyzed (Participants) | 68 | 67 | 67 | 69
  Sodium: Follow up | 0.1 (2.3) | -0.3 (1.7) | 0.6 (1.8) | 0.2 (1.9)
  Potassium: 24 hour post dose | 0.26 (0.41) | 0.25 (0.39) | 0.17 (0.41) | 0.11 (0.36)
  Potassium: Follow up: number analyzed (Participants) | 68 | 67 | 67 | 69
  Potassium: Follow up | 0.01 (0.33) | -0.02 (0.45) | 0.01 (0.40) | -0.01 (0.41)
  Chloride: 24 hour post dose | 1.3 (2.0) | 1.0 (1.9) | 1.4 (2.0) | 1.4 (2.0)
  Chloride: Follow up: number analyzed (Participants) | 68 | 67 | 67 | 69
  Chloride: Follow up | 0.3 (2.1) | -0.3 (2.3) | 0.5 (1.7) | 0.1 (2.1)
  Bicarbonate: 24 hour post dose | 0.2 (2.4) | 0.1 (1.8) | 0.6 (1.9) | 0.4 (2.1)
  Bicarbonate: Follow up: number analyzed (Participants) | 68 | 67 | 67 | 69
  Bicarbonate: Follow up | -0.2 (2.2) | -0.3 (2.2) | 0.3 (2.1) | -0.1 (2.2)

30. Secondary Outcome: Changes From Baseline for Magnesium, Glucose (Fasting), Blood Urea Nitrogen (BUN), Creatinine, Total Bilirubin, Direct Bilirubin
Description: Change from baseline calculated by subtracting the Day -1 (baseline) chemistry measurement from the 24 h post dose, and a follow up chemistry measurement. Follow up is defined as either the check-in visit for the next period or the final visit. Chemistry parameters included magnesium, glucose (fasting), BUN, creatinine, total bilirubin, direct bilirubin
Time Frame: Prior to dosing, 24 hour post dose through prior to the next dose (Day 8 or Final visit).
Population: Any participants who received study product for that dosing period and had post dose laboratory assessments.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | 2 g of Zoliflodacin | 4 g of Zoliflodacin | Placebo | 400 mg of Moxifloxacin
Number analyzed (Participants) | 69 | 67 | 70 | 70
mg/dL
  Magnesium: 24 hour post dose | 0.05 (0.13) | 0.03 (0.13) | 0.02 (0.14) | 0.01 (0.14)
  Magnesium: Follow up: number analyzed (Participants) | 68 | 67 | 67 | 69
  Magnesium: Follow up | 0.04 (0.12) | 0.00 (0.13) | 0.02 (0.13) | 0.01 (0.12)
  Glucose (fasting): 24 hour post dose: number analyzed (Participants) | 69 | 67 | 69 | 67
  Glucose (fasting): 24 hour post dose | 4.6 (7.8) | 6.4 (9.7) | 4.2 (8.3) | 3.2 (7.4)
  Glucose (fasting): Follow up: number analyzed (Participants) | 67 | 67 | 66 | 66
  Glucose (fasting): Follow up | -1.2 (8.7) | 1.5 (9.8) | -0.6 (8.9) | 1.0 (9.5)
  BUN: 24 hour post dose | 2.1 (3.2) | 1.6 (3.0) | 1.4 (2.9) | 2.5 (3.4)
  BUN: Follow up: number analyzed (Participants) | 68 | 67 | 67 | 69
  BUN: Follow up | 0.7 (3.3) | 0.0 (2.9) | 0.1 (3.0) | -0.2 (4.0)
  Creatinine: 24 hour post dose | 0.082 (0.082) | 0.086 (0.072) | 0.003 (0.059) | 0.059 (0.078)
  Creatinine: Follow up: number analyzed (Participants) | 68 | 67 | 67 | 69
  Creatinine: Follow up | 0.034 (0.102) | -0.011 (0.089) | 0.006 (0.071) | -0.007 (0.087)
  Total Bilirubin: 24 hour post dose | 0.07 (0.25) | 0.14 (0.23) | -0.01 (0.24) | -0.04 (0.20)
  Total Bilirubin: Follow up: number analyzed (Participants) | 68 | 67 | 67 | 69
  Total Bilirubin: Follow up | 0.01 (0.21) | -0.04 (0.14) | -0.01 (0.17) | -0.02 (0.16)
  Direct Bilirubin: 24 hour post dose | 0.00 (0.07) | 0.02 (0.06) | 0.00 (0.06) | -0.01 (0.05)
  Direct Bilirubin: Follow up: number analyzed (Participants) | 68 | 66 | 67 | 69
  Direct Bilirubin: Follow up | -0.01 (0.06) | 0.00 (0.05) | 0.01 (0.06) | -0.01 (0.05)

31. Secondary Outcome: Changes From Baseline for Total Protein and Albumin
Description: Change from baseline calculated by subtracting the Day -1 (baseline) chemistry measurement from the 24 h post dose, and a follow up chemistry measurement. Follow up is defined as either the check-in visit for the next period or the final visit. Chemistry parameters included total protein and albumin.
Time Frame: Prior to dosing, 24 hour post dose through prior to the next dose (Day 8 or Final visit).
Population: Any participants who received study product for that dosing period and had post dose laboratory assessments.
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | 2 g of Zoliflodacin | 4 g of Zoliflodacin | Placebo | 400 mg of Moxifloxacin
Number analyzed (Participants) | 69 | 67 | 70 | 70
g/dL
  Total Protein: 24 hour post dose | -0.42 (0.45) | -0.42 (0.39) | -0.45 (0.43) | -0.45 (0.38)
  Total Protein: Follow up: number analyzed (Participants) | 68 | 67 | 67 | 69
  Total Protein: Follow up | -0.01 (0.49) | -0.06 (0.39) | -0.01 (0.40) | 0.03 (0.41)
  Albumin: 24 hour post dose | -0.28 (0.25) | -0.30 (0.23) | -0.30 (0.24) | -0.32 (0.23)
  Albumin: Follow up: number analyzed (Participants) | 68 | 67 | 67 | 69
  Albumin: Follow up | 0.00 (0.28) | -0.05 (0.22) | 0.01 (0.23) | 0.02 (0.23)

32. Secondary Outcome: Changes From Baseline for Aspartate Aminotransferase (AST), Alanine Aminotransferase (ALT) and Alkaline Phosphatase (AP)
Description: Change from baseline calculated by subtracting the Day -1 (baseline) chemistry measurement from the 24 h post dose, and a follow up chemistry measurement. Follow up is defined as either the check-in visit for the next period or the final visit. Chemistry parameters included AST, ALT and AP.
Time Frame: Prior to dosing, 24 hour post dose through prior to the next dose (Day 8 or Final visit).
Population: Any participants who received study product for that dosing period and had post dose laboratory assessments.
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | 2 g of Zoliflodacin | 4 g of Zoliflodacin | Placebo | 400 mg of Moxifloxacin
Number analyzed (Participants) | 69 | 67 | 70 | 70
U/L
  AST: 24 hour post dose | -2.9 (3.0) | -2.7 (5.6) | -2.7 (3.5) | -2.8 (4.4)
  AST: Follow up: number analyzed (Participants) | 68 | 67 | 67 | 69
  AST: Follow up | 0.1 (5.6) | 0.0 (4.0) | -0.5 (3.3) | 0.6 (5.9)
  ALT: 24 hour post dose | -2.2 (4.1) | -1.7 (2.7) | -1.7 (4.0) | -1.4 (3.8)
  ALT: Follow up: number analyzed (Participants) | 68 | 67 | 67 | 69
  ALT: Follow up | -0.7 (6.9) | 1.6 (7.5) | -0.6 (4.2) | 0.8 (4.3)
  AP: 24 hour post dose | -5.2 (6.3) | -3.9 (4.6) | -4.1 (4.9) | -4.2 (5.8)
  AP: Follow up: number analyzed (Participants) | 68 | 67 | 67 | 69
  AP: Follow up | -1.7 (8.1) | -0.4 (7.0) | -0.7 (4.8) | 1.0 (7.0)

33. Secondary Outcome: Changes From Baseline for Glomerular Filtration Rate (GFR) - Estimated
Description: Change from baseline calculated by subtracting the Day -1 (baseline) chemistry measurement from the 24 h post dose, and a follow up chemistry measurement. Follow up is defined as either the check-in visit for the next period or the final visit.
Time Frame: Prior to dosing, 24 hour post dose through prior to the next dose (Day 8 or Final visit).
Population: Any participants who received study product and had post dose laboratory assessments.
Measure: Mean (Standard Deviation); unit: mL/minute
Arm/Group | 2 g of Zoliflodacin | 4 g of Zoliflodacin | Placebo | 400 mg of Moxifloxacin
Number analyzed (Participants) | 69 | 67 | 70 | 70
mL/minute
  GFR: 24 hour post dose | -10.4 (11.1) | -9.5 (8.1) | -0.1 (8.1) | -6.2 (10.3)
  GFR: Follow up: number analyzed (Participants) | 68 | 67 | 67 | 69
  GFR: Follow up | -5.3 (16.3) | 1.8 (11.0) | -0.7 (8.5) | 1.5 (11.9)

34. Secondary Outcome: Occurrence of Urinalysis Adverse Events Following Administration of Study Product
Description: Urine for the clinical laboratory test was collected on Day -1, 24 hour post dose and the check in for the following dosing period. The results for glucose dipstick, protein dipstick and occult blood - dipstick were reported in categorical results. The possibilities were negative, trace, 1+, 2+, and 3+. If the dipsticks were 1+ or greater, microscopic evaluations were performed for erythrocytes, leukocytes and bacteria. For microscopic results to be deemed abnormal, the results must be reported 6 or greater per high power field.
Time Frame: From study product administration (Day 1) through prior to the next dose (Day 8 or Final visit).
Population: Any participants who received study product and had post dose laboratory assessments.
Measure: Count of Participants; unit: Participants
Arm/Group | 2 g of Zoliflodacin | 4 g of Zoliflodacin | Placebo | 400 mg of Moxifloxacin
Number analyzed (Participants) | 69 | 67 | 70 | 70
Participants
  Glucose dipstick: 24 hour post dose | 0 | 0 | 0 | 0
  Glucose dipstick: Follow up: number analyzed (Participants) | 68 | 67 | 67 | 69
  Glucose dipstick: Follow up | 0 | 0 | 0 | 0
  Protein dipstick: 24 hour post dose | 1 | 1 | 0 | 0
  Protein dipstick: Follow up: number analyzed (Participants) | 68 | 67 | 67 | 69
  Protein dipstick: Follow up | 2 | 0 | 0 | 1
  Occult blood dipstick: 24 hour post dose | 1 | 4 | 5 | 3
  Occult blood dipstick: Follow up: number analyzed (Participants) | 68 | 67 | 67 | 69
  Occult blood dipstick: Follow up | 4 | 2 | 0 | 1
  Erythrocytes microscopic: 24 hour post dose: number analyzed (Participants) | 69 | 67 | 68 | 70
  Erythrocytes microscopic: 24 hour post dose | 2 | 2 | 2 | 3
  Erythrocytes microscopic: Follow up: number analyzed (Participants) | 68 | 67 | 67 | 69
  Erythrocytes microscopic: Follow up | 3 | 1 | 2 | 2
  Leukocytes microscopic: 24 hour post dose: number analyzed (Participants) | 69 | 67 | 68 | 70
  Leukocytes microscopic: 24 hour post dose | 0 | 1 | 0 | 2
  Leukocytes microscopic: Follow up: number analyzed (Participants) | 68 | 67 | 67 | 69
  Leukocytes microscopic: Follow up | 0 | 0 | 1 | 0
  Bacteria microscopic: 24 hour post dose: number analyzed (Participants) | 69 | 67 | 68 | 70
  Bacteria microscopic: 24 hour post dose | 0 | 3 | 2 | 2
  Bacteria microscopic: Follow up: number analyzed (Participants) | 68 | 67 | 67 | 69
  Bacteria microscopic: Follow up | 2 | 1 | 2 | 0

35. Secondary Outcome: Changes From Baseline in ECG Measures: PR Interval, QRS Duration, QT Interval, QTcF Interval and RR Interval
Description: Change from baseline in ECG is calculated by subtracting the baseline (pre-dose) measurement from the post-dose measurement. Post-dose measurements were taken 1 h, 2 h, 4 h, 24 h after dosing and prior to the next dose (follow up). The following ECG Parameters were analyzed: PR Interval (Interval From Onset of P-wave to the Onset of the QRS Complex), QRS Duration (Time From the Start of the Q-wave to the End of the S-wave), QT Interval (Interval From Onset of the Q-wave to the End of the T-wave), QTcF Interval (QT Interval Corrected by Fridericia's Formula) and RR Interval (Interval From the Peak of the R Wave of a QRS Complex to the Peak of the R Wave of the Next QRS Complex).
Time Frame: Baseline, 1 h, 2 h, 4h, 24 h post-dose and follow up
Population: Any participants who received study product and had post dose ECG assessments.
Measure: Mean (Standard Deviation); unit: milliseconds (msec)
Arm/Group | 2 g of Zoliflodacin | 4 g of Zoliflodacin | Placebo | 400 mg of Moxifloxacin
Number analyzed (Participants) | 69 | 67 | 70 | 71
milliseconds (msec)
  PR Interval: 1 hr post dose | 1.2 (8.9) | 0.0 (7.7) | 1.3 (8.5) | 1.3 (11.7)
  PR Interval: 2 hr post dose | 1.2 (8.3) | -0.7 (7.8) | 0.6 (7.6) | 0.4 (11.5)
  PR Interval: 4 hr post dose: number analyzed (Participants) | 69 | 67 | 70 | 70
  PR Interval: 4 hr post dose | -0.3 (8.0) | -1.4 (8.3) | -0.4 (7.8) | -0.9 (11.6)
  PR Interval: 24 hr post dose: number analyzed (Participants) | 69 | 67 | 70 | 70
  PR Interval: 24 hr post dose | 1.1 (7.8) | 0.7 (7.9) | 0.5 (8.2) | 2.8 (11.3)
  PR Interval: Follow up: number analyzed (Participants) | 68 | 67 | 67 | 69
  PR Interval: Follow up | -1.2 (8.8) | -1.9 (9.8) | -3.1 (9.9) | -0.9 (13.3)
  QRS Duration: 1 hr post dose | -1.8 (4.1) | -0.6 (5.1) | 0.4 (5.1) | -0.5 (6.7)
  QRS Duration: 2 hr post dose | -1.9 (6.6) | -1.4 (4.9) | -0.7 (5.9) | -1.5 (8.0)
  QRS Duration: 4 hr post dose: number analyzed (Participants) | 69 | 67 | 70 | 70
  QRS Duration: 4 hr post dose | -2.0 (3.9) | -1.0 (5.2) | -0.7 (5.1) | -1.6 (7.4)
  QRS Duration: 24 hr post dose: number analyzed (Participants) | 69 | 67 | 70 | 70
  QRS Duration: 24 hr post dose | -2.7 (4.9) | -1.1 (6.8) | -0.9 (5.0) | -1.1 (7.0)
  QRS Duration: Follow up: number analyzed (Participants) | 68 | 67 | 67 | 69
  QRS Duration: Follow up | -1.4 (6.0) | 0.3 (6.9) | -1.1 (5.3) | -0.2 (8.6)
  QT Interval: 1 hr post dose | -3.6 (13.1) | -6.2 (12.2) | -2.5 (11.1) | -1.4 (12.6)
  QT Interval: 2 hr post dose | -5.3 (14.6) | -7.6 (15.6) | -3.6 (13.3) | 2.3 (16.7)
  QT Interval: 4 hr post dose: number analyzed (Participants) | 69 | 67 | 70 | 70
  QT Interval: 4 hr post dose | -5.0 (13.8) | -9.1 (18.3) | -3.8 (14.3) | 2.0 (16.1)
  QT Interval: 24 hr post dose: number analyzed (Participants) | 69 | 67 | 70 | 70
  QT Interval: 24 hr post dose | -6.8 (12.3) | -7.6 (15.9) | -9.9 (15.1) | -3.7 (14.1)
  QT Interval: Follow up: number analyzed (Participants) | 68 | 67 | 67 | 69
  QT Interval: Follow up | -7.1 (20.7) | -6.6 (21.1) | -8.3 (20.2) | -10.0 (18.4)
  QTcF Interval: 1 hr post dose | 1.5 (10.8) | 0.6 (9.3) | -0.4 (9.2) | 9.2 (10.9)
  QTcF Interval: 2 hr post dose | 0.4 (9.9) | 2.0 (10.2) | -2.9 (9.5) | 10.6 (11.5)
  QTcF Interval: 4 hr post dose: number analyzed (Participants) | 69 | 67 | 70 | 70
  QTcF Interval: 4 hr post dose | 0.7 (10.8) | -1.3 (12.2) | -3.0 (9.9) | 8.5 (12.0)
  QTcF Interval: 24 hr post dose: number analyzed (Participants) | 69 | 67 | 70 | 70
  QTcF Interval: 24 hr post dose | 1.5 (8.5) | 1.9 (9.3) | -3.5 (10.3) | 4.1 (11.6)
  QTcF Interval: Follow up: number analyzed (Participants) | 68 | 67 | 67 | 69
  QTcF Interval: Follow up | -1.4 (12.7) | -0.2 (12.8) | -3.8 (14.4) | -1.4 (14.9)
  RR Interval: 1 hr post dose | -34.9 (99.9) | -48.4 (86.0) | -14.1 (80.6) | -74.5 (100.2)
  RR Interval: 2 hr post dose | -38.5 (99.7) | -68.7 (82.0) | -3.3 (94.0) | -59.0 (107.3)
  RR Interval: 4 hr post dose: number analyzed (Participants) | 69 | 67 | 70 | 70
  RR Interval: 4 hr post dose | -38.8 (94.7) | -54.3 (102.3) | -4.8 (113.1) | -46.6 (114.0)
  RR Interval: 24 hr post dose: number analyzed (Participants) | 69 | 67 | 70 | 70
  RR Interval: 24 hr post dose | -57.6 (83.5) | -66.9 (91.3) | -45.9 (106.1) | -56.8 (87.0)
  RR Interval: Follow up: number analyzed (Participants) | 68 | 67 | 67 | 69
  RR Interval: Follow up | -39.6 (112.7) | -45.6 (108.6) | -32.4 (125.5) | -62.1 (103.1)

36. Secondary Outcome: Changes From Baseline in ECG Measures: Ventricular Rate
Description: Change from baseline in ECG Ventricular Rate is calculated by subtracting the baseline (pre-dose) measurement from the post-dose measurement. Post-dose measurements were taken 1 h, 2 h, 4 h, 24 h after dosing and prior to the next dose (follow up).
Time Frame: Baseline, 1 h, 2 h, 4h, 24 h post-dose and follow up
Population: Any participants who received study product and had post dose ECG assessments.
Measure: Mean (Standard Deviation); unit: beats/minute
Arm/Group | 2 g of Zoliflodacin | 4 g of Zoliflodacin | Placebo | 400 mg of Moxifloxacin
Number analyzed (Participants) | 69 | 67 | 70 | 71
beats/minute
  Ventricular Rate: 1 hr post dose | 2.4 (6.6) | 3.3 (5.3) | 0.9 (5.1) | 4.7 (6.2)
  Ventricular Rate: 2 hr post dose | 2.9 (6.8) | 4.6 (6.2) | 0.4 (6.5) | 3.6 (6.8)
  Ventricular Rate: 4 hr post dose: number analyzed (Participants) | 69 | 67 | 70 | 70
  Ventricular Rate: 4 hr post dose | 2.8 (6.6) | 4.1 (7.5) | 0.2 (7.3) | 2.8 (7.4)
  Ventricular Rate: 24 hr post dose: number analyzed (Participants) | 69 | 67 | 70 | 70
  Ventricular Rate: 24 hr post dose | 3.9 (5.8) | 4.6 (6.4) | 2.9 (8.0) | 3.5 (5.8)
  Ventricular Rate: Follow up: number analyzed (Participants) | 68 | 67 | 67 | 69
  Ventricular Rate: Follow up | 2.8 (8.2) | 3.1 (7.3) | 1.8 (8.9) | 3.9 (7.0)

ADVERSE EVENTS:
Time Frame: Unsolicited adverse events and serious adverse events (SAEs) were collected from study product administration to Day 8 after treatment administration or final visit.
Description: Treatment emergent adverse events were defined as new events post-dose, or worsening of existing conditions post-dose. The adverse events were captured by changes in laboratory values, vital signs, ECGs and unsolicited adverse events immediately post dose to Day 8 post each treatment administration or early termination, whichever came first.
Arm/Group | 2 g of Zoliflodacin | 4 g of Zoliflodacin | Placebo | 400 mg of Moxifloxacin
All-Cause Mortality (participants affected / at risk) | 0/69 | 0/67 | 0/70 | 0/71
Serious Adverse Events (participants affected / at risk) | 0/69 | 0/67 | 0/70 | 0/71
Other Adverse Events (participants affected / at risk) | 38/69 | 46/67 | 30/70 | 34/71
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 2 g of Zoliflodacin (N=69) | 4 g of Zoliflodacin (N=67) | Placebo (N=70) | 400 mg of Moxifloxacin (N=71)
DIARRHOEA (Gastrointestinal disorders) | 0 (0) | 4 (4) | 0 (0) | 0 (0)
NAUSEA (Gastrointestinal disorders) | 2 (2) | 6 (6) | 1 (1) | 3 (3)
BACTERIAL TEST POSITIVE (Investigations) | 2 (2) | 4 (4) | 5 (5) | 2 (2)
ELECTROCARDIOGRAM QT PROLONGED (Investigations) | 5 (8) | 3 (4) | 2 (2) | 15 (15)
HAEMOGLOBIN DECREASED (Investigations) | 2 (2) | 4 (4) | 3 (3) | 1 (1)
HEART RATE DECREASED (Investigations) | 13 (14) | 10 (12) | 13 (16) | 11 (16)
NEUTROPHIL COUNT DECREASED (Investigations) | 1 (1) | 4 (4) | 2 (2) | 1 (1)
DYSGEUSIA (Nervous system disorders) | 6 (6) | 5 (5) | 2 (2) | 0 (0)
HEADACHE (Nervous system disorders) | 7 (7) | 12 (13) | 2 (2) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2018-11-27): https://cdn.clinicaltrials.gov/large-docs/49/NCT03613649/Prot_000.pdf
  • Statistical Analysis Plan (2018-12-19): https://cdn.clinicaltrials.gov/large-docs/49/NCT03613649/SAP_001.pdf